CLINICAL TRIAL: NCT01751906
Title: A Clinical Evaluation of Absorb™ BVS, the Everolimus Eluting Bioresorbable Vascular Scaffold in the Treatment of Subjects With de Novo Native Coronary Artery Lesions.
Brief Title: ABSORB III Randomized Controlled Trial (RCT)
Acronym: ABSORB-III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-392
Record Dates: First submitted 2012-12-13; First posted 2012-12-18 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease; Coronary Artery Stenosis; Coronary Disease; Coronary Stenosis
Keywords: Absorb™ BVS; Angioplasty; Bioabsorbable; BVS; Bioresorbable; Coronary Artery Disease; Coronary Artery Endothelial Responsiveness; Coronary artery restenosis; Coronary artery stenosis; Coronary scaffold; Coronary Stent; Drug eluting stents; Everolimus; Myocardial ischemia; Stent thrombosis; Stents
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Coronary Disease; Coronary Restenosis; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Absorb BVS (Experimental): Subjects receiving Absorb BVS
  Interventions: Device: Absorb BVS
- XIENCE (Active Comparator): Subjects receiving XIENCE V, XIENCE PRIME, or XIENCE Xpedition
  Interventions: Device: XIENCE

INTERVENTIONS:
Device: Absorb BVS — * Scaffold diameters: 2.5, 3.0 and 3.5 mm
  * Scaffold lengths: 8, 12, 18, and 28 mm The 3.0 x 18 mm Absorb BVS will be used for the Lead-In. Both the 8 mm and 12 mm lengths will be available for the 2.5/3.0 mm diameter Absorb BVS. Only the 12 mm length will be available for the 3.5 mm diameter.
  * The commercially approved CE marked device will be used in geographies where it is commercially available. The commercially approved CE marked 23mm Absorb BVS device will not be used in this study.
  Bioabsorbable drug eluting stent implantation for improving coronary luminal diameter in patients, including those with diabetes mellitus, with ischemic heart disease due to de novo native coronary artery lesions (length ≤ 24 mm) with a reference vessel diameter of ≥ 2.5 mm and ≤ 3.75 mm.
  Arms: Absorb BVS
Device: XIENCE — Commercially approved XIENCE Family Stent System, inclusive of XIENCE V, XIENCE PRIME, XIENCE Xpedition, XIENCE Alpine, XIENCE Pro (OUS only), and XIENCE ProX (OUS only).
  * Stent diameters: 2.5, 2.75, 3.0, 3.25, 3.5 and 4.0 mm
  * Stent lengths: 8, 12, 15, 18, 23, and 28 mm. The 3.25 mm is only available for XIENCE Xpedition
  * For geographies where these devices are commercially available, the investigational sties may use only their locally approved devices
  To improve coronary luminal diameter in patients, including those with diabetes mellitus, with ischemic heart disease due to de novo native coronary artery lesions (length ≤ 24 mm) with a reference vessel diameter of ≥ 2.5 mm and ≤ 3.75 mm.
  Arms: XIENCE

SUMMARY:
The ABSORB III RCT is a prospective randomized, single-blind, multi-center trial. It is the pivotal trial to support the US pre-market approval (PMA) of Absorb™ Bioresorbable Vascular Scaffold (BVS).

The ABSORB III includes additional two trials i.e. ABSORB III PK (pharmacokinetics) sub-study and ABSORB IV RCT trial which are maintained under one protocol because both trial designs are related, ABSORB IV is the continuation of ABSORB III and the data from ABSORB III and ABSORB IV will be pooled to support the ABSORB IV primary endpoint. Both the trials will evaluate the safety and effectiveness of Absorb BVS.

DETAILED DESCRIPTION:
ABSORB III RCT:

A. Primary Objective: The pivotal trial to support the US pre-market approval (PMA) of Absorb BVS. ABSORB III will evaluate the safety and effectiveness of the Absorb BVS System compared to the XIENCE in the treatment of subjects, including those with diabetes mellitus, with ischemic heart disease caused by up to two de novo native coronary artery lesions in separate epicardial vessels.

B. Powered Secondary Objectives:

1. Lead-In Phase Objective: To evaluate the applicability and transferability of the didactic Absorb BVS physician training plan to US clinical practice.

   The lead-in phase is a non-randomized, single-arm, open label group of up to 50 subjects treated with Absorb BVS at up to 35 US sites. The Lead-In phase will enroll/register subjects prior to the randomization phase of ABSORB III.

   The Lead-In Phase allows the treatment of up to two de novo native coronary artery lesions in different epicardial vessels with reference vessel diameter (RVD) ≥ 2.75 mm to ≤ 3.25 mm and lesion lengths ≥ 8 to ≤ 14 mm.
2. Imaging Cohort Objective: To evaluate long-term vascular function and patency of the Absorb BVS treated segments compared to XIENCE treated segments in the treatment of subjects with ischemic heart disease caused by up to two de novo native coronary artery lesions in separate epicardial vessels.

The imaging cohort-phase is a prospective, randomized (2:1 Absorb BVS to XIENCE), single-blind, multi-center trial, registering approximately 200 subjects. This includes 150 subjects for the angiographic/intravascular ultrasound (IVUS) endpoints analysis and approximately 50 subjects for optical coherence tomography (OCT) endpoints analysis. The 200 subjects are separate from the 2000 subjects included in the primary analysis. Data from two powered secondary endpoints from this cohort will support label claims of superiority of Absorb BVS as compared to XIENCE specific to vasomotion and late lumen enlargement.

All other subjects in ABSORB III unless specified will receive treatment of up to two de novo native coronary artery lesions in different epicardial vessels with RVD ≥ 2.5 mm to ≤ 3.75 mm and lesion lengths ≤ 24 mm.

ELIGIBILITY:
General Inclusion Criteria:

1. Subject must be at least 18 years of age.
2. Subject or a legally authorized representative must provide written Informed Consent prior to any study related procedure, per site requirements.
3. Subject must have evidence of myocardial ischemia (e.g., stable, unstable angina, post-infarct angina or silent ischemia) suitable for elective PCI. Subjects with stable angina or silent ischemia and < 70% diameter stenosis must have objectives sign of ischemia as determined by one of the following, echocardiogram, nuclear scan, ambulatory ECG or stress ECG). In the absence of noninvasive ischemia, fractional flow reserve (FFR) must be done and indicative of ischemia.
4. Subject must be an acceptable candidate for coronary artery bypass graft (CABG) surgery.
5. Female subject of childbearing potential who does not plan pregnancy for up to 1 year following the index procedure. For a female subject of childbearing potential a pregnancy test must be performed with negative results known within 7 days prior to the index procedure per site standard.
6. Female subject is not breast-feeding at the time of the screening visit and will not be breast-feeding for up to 1 year following the index procedure.
7. Subject agrees to not participate in any other investigational or invasive clinical study for a period of 1 year following the index procedure.

Angiographic Inclusion Criteria:

1. One or two de novo target lesions:

   1. If there is one target lesion, a second non-target lesion may be treated but the non-target lesion must be present in a different epicardial vessel, and must be treated first with a successful, uncomplicated result prior to randomization of the target lesion.
   2. If two target lesions are present, they must be present in different epicardial vessels and both must satisfy the angiographic eligibility criteria.
   3. The definition of epicardial vessels means the LAD, LCX and RCA and their branches. Thus, the patient must not have lesions requiring treatment in e.g. both the LAD and a diagonal branch.
2. Target lesion(s) must be located in a native coronary artery with a visually estimated or quantitatively assessed %DS of ≥ 50% and < 100% with a TIMI flow of ≥ 1 and one of the following: stenosis ≥ 70%, an abnormal functional test (e.g., fractional flow reserve, stress test), unstable angina or post-infarct angina.

   1. Lesion(s) must be located in a native coronary artery with RVD by visual estimation of ≥ 2.50 mm and ≤ 3.75 mm.
   2. Lesion(s) must be located in a native coronary artery with length by visual estimation of ≤ 24 mm.
   3. For Lead-In subjects with 3.0x18 mm Absorb BVS: lesions (s) must be located in a native coronary artery with RVD by visual estimation of ≥ 2.75 mm and ≤ 3.25 mm. The lesion length by visual estimation is ≥ 8 mm and ≤ 14 mm.

General Exclusion Criteria:

1. Any surgery requiring general anesthesia or discontinuation of aspirin and/or an ADP antagonist is planned within 12 months after the procedure.
2. Subject has known hypersensitivity or contraindication to device material and its degradants (everolimus, poly (L-lactide), poly (DL-lactide), lactide, lactic acid) and cobalt, chromium, nickel, platinum, tungsten, acrylic and fluoro polymers that cannot be adequately pre-medicated. Subject has a known contrast sensitivity that cannot be adequately pre-medicated.
3. Subject has known allergic reaction, hypersensitivity or contraindication to aspirin; or to clopidogrel and prasugrel and ticagrelor; or to heparin and bivalirudin, and therefore cannot be adequately treated with study medications.
4. Subject had an acute myocardial infarction (AMI; STEMI or NSTEMI) within 72 hours of the index procedure and both CK and CK-MB have not returned to within normal limits at the time of index procedure; or subject with stable angina or silent ischemia has CK-MB that is greater than normal limits at the time of the index procedure.
5. Subject is currently experiencing clinical symptoms consistent with new onset AMI (STEMI or NSTEMI), such as nitrate-unresponsive prolonged chest pain with ischemic ECG changes.
6. Subject has a cardiac arrhythmia as identified at the time of screening for which at least one of the following criteria is met:

   1. Subject requires coumadin or any other agent for chronic oral anticoagulation.
   2. Subject is likely to become hemodynamically unstable due to their arrhythmia.
   3. Subject has poor survival prognosis due to their arrhythmia.
7. Subject has a left ventricular ejection fraction (LVEF) < 30% assessed by any quantitative method, including but not limited to echocardiography, MRI, Multiple-Gated Acquisition (MUGA) scan, contrast left ventriculography, PET scan, etc. LVEF may be obtained within 6 months prior to the procedure for subjects with stable CAD. For subjects presenting with ACS, LVEF must be assessed during the index hospitalization (which may include during the index procedure by contrast left ventriculography) but prior to randomization in order to confirm the subject's eligibility.
8. Subject has undergone prior PCI within the target vessel during the last 12 months. Prior PCI within the non-target vessel or any peripheral intervention is acceptable if performed anytime >30 days before the index procedure, or between 24 hours and 30 days before the index procedure if successful and uncomplicated.
9. Subject requires future staged PCI either in target or non-target vessels or subject requires future peripheral interventions < 30 days after the index procedure
10. Subject has received any solid organ transplants or is on a waiting list for any solid organ transplants.
11. At the time of screening, the subject has a malignancy that is not in remission.
12. Subject is receiving immunosuppressant therapy or has known immunosuppressive or severe autoimmune disease that requires chronic immunosuppressive therapy (e.g., human immunodeficiency virus, systemic lupus erythematosus, etc.). Note: corticosteroids are not included as immunosuppressant therapy.
13. Subject has previously received or is scheduled to receive radiotherapy to a coronary artery (vascular brachytherapy), or the chest/mediastinum.
14. Subject is receiving or will require chronic anticoagulation therapy (e.g., coumadin, dabigatran, apixaban, rivaroxaban or any other agent for any reason).
15. Subject has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3.
16. Subject has a documented or suspected hepatic disorder as defined as cirrhosis or Child-Pugh ≥ Class B.
17. Subject has renal insufficiency as defined as an estimated GFR < 30 ml/min/1.73m2 or dialysis at the time of screening.
18. Subject is high risk of bleeding for any reason; has a history of bleeding diathesis or coagulopathy; has had a significant gastro-intestinal or significant urinary bleed within the past six months.
19. Subject has had a cerebrovascular accident or transient ischemic neurological attack (TIA) within the past six months, or any prior intracranial bleed, or any permanent neurologic defect, or any known intracranial pathology (e.g. aneurysm, arteriovenous malformation, etc.).
20. Subject has extensive peripheral vascular disease that precludes safe 6 French sheath insertion. Note: femoral arterial disease does not exclude the patient if radial access may be used.
21. Subject has life expectancy < 5 years for any non-cardiac cause or cardiac cause.
22. Subject is in the opinion of the Investigator or designee, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason. This includes completion of Patient Reported Outcome instruments.
23. Subject is currently participating in another clinical trial that has not yet completed its primary endpoint.
24. Subject is part of a vulnerable population who, in the judgment of the investigator, is unable to give Informed Consent for reasons of incapacity, immaturity, adverse personal circumstances or lack of autonomy. This may include: Individuals with mental disability, persons in nursing homes, children, impoverished persons, persons in emergency situations, homeless persons, nomads, refugees, and those incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention.

Angiographic Exclusion Criteria:

All exclusion criteria apply to the target lesion(s) or target vessel(s).

1. Lesion which prevents successful balloon pre-dilatation, defined as full balloon expansion with the following outcomes:

   1. Residual %DS is a maximum < 40% (per visual estimation), ≤ 20% is strongly recommended.
   2. TIMI Grade-3 flow (per visual estimation).
   3. No angiographic complications (e.g. distal embolization, side branch closure).
   4. No dissections NHLBI grade D-F.
   5. No chest pain lasting > 5 minutes.
   6. No ST depression or elevation lasting > 5 minutes.
2. Lesion is located in left main.
3. Aorto-ostial RCA lesion (within 3 mm of the ostium).
4. Lesion located within 3 mm of the origin of the LAD or LCX.
5. Lesion involving a bifurcation with a:

   1. side branch ≥ 2 mm in diameter, or
   2. side branch with either an ostial or non-ostial lesion with diameter stenosis > 50%, or
   3. side branch requiring dilatation
6. Anatomy proximal to or within the lesion that may impair delivery of the Absorb BVS or XIENCE stent:

   1. Extreme angulation (≥ 90°) proximal to or within the target lesion.
   2. Excessive tortuosity (≥ two 45° angles) proximal to or within the target lesion.
   3. Moderate or heavy calcification proximal to or within the target lesion. If IVUS used, subject must be excluded if calcium arc in the vessel prior to the lesion or within the lesion is ≥ 180°.
7. Vessel contains thrombus as indicated in the angiographic images or by IVUS or OCT.
8. Lesion or vessel involves a myocardial bridge.
9. Vessel has been previously treated with a stent at any time prior to the index procedure such that the Absorb BVS or XIENCE would need to cross the stent to reach the target lesion.
10. Vessel has been previously treated and the target lesion is within 5 mm proximal or distal to a previously treated lesion.
11. Target lesion located within an arterial or saphenous vein graft or distal to any arterial or saphenous vein graft.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2008 (Actual)
Dates: Start 2012-12; Primary Completion 2016-09 (Actual); Study Completion 2020-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen G Ellis, MD, Principal Investigator — Cleveland Clinic, Cleveland OH; Dean J Kereiakes, MD, Principal Investigator — The Christ Hospital, Cincinnati, OH; Gregg W Stone, MD, Study Chair — Columbia University Medical Center, New York, NY; Jennifer McMeans Jones, Study Director — Abbott Medical Devices
Locations (192):
- United States (190):
  - Baptist Medical Center Princeton, Birmingham, Alabama
  - University of Alabama Hospital, Birmingham, Alabama
  - Thomas Hospital, Fairhope, Alabama
  - Baptist Medical Center South, Montgomery, Alabama
  - Chandler Regional Medical Center, Gilbert, Arizona
  - Banner Heart Hospital, Mesa, Arizona
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - John Muir Medical Center - Concord Campus, Concord, California
  - Washington Hospital, Fremont, California
  - Scripps Green Hospital, La Jolla, California
  - Scripps Memorial Hospital, La Jolla, California
  - Good Samaritan Hospital, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Sutter Central Valley Hospitals dba Memorial Medical Center, Modesto, California
  - Mercy General Hospital, Sacramento, California
  - UC Davis Medical Center, Sacramento, California
  - Sutter Medical Center, Sacramento, California
  - Sharp Memorial Hospital, San Diego, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Stanford Hospital and Clinics, Stanford, California
  - Little Company Of Mary Hospital, Torrance, California
  - Torrance Memorial Medical Center, Torrance, California
  - UCH-Memorial Health Systems, Colorado Springs, Colorado
  - Medical Center of the Rockies, Fort Collins, Colorado
  - Yale-New Haven Hospital, New Haven, Connecticut
  - St. Vincent's Medical Center, Stamford, Connecticut
  - Christiana Care Health Services, Newark, Delaware
  - Brandon Regional Hospital, Brandon, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - St. Vincent's Medical Center, Jacksonville, Florida
  - Baptist Medical Center - Downtown, Jacksonville, Florida
  - University of Florida UF Health, Jacksonville, Florida
  - University of Miami Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - MediQuest Research Group Inc at Munroe Regional Medical Center, Ocala, Florida
  - Florida Hospital, Orlando, Florida
  - Palm Beach Gardens Medical Center, Palm Beach Gardens, Florida
  - Bay County Health Systems, Panama City, Florida
  - Baptist Hospital, Pensacola, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Tampa General Hospital, Tampa, Florida
  - Florida Hospital Pepin Heart Institute, Tampa, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - University Hospital, Augusta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Saint Francis Medical Center, Peoria, Illinois
  - St. John's Hospital, Springfield, Illinois
  - Elkhart General Healthcare, Elkhart, Indiana
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Genesis Medical Center, Davenport, Iowa
  - Mercy Medical, West Des Moines, Iowa
  - The University of Kansas Hospital and Medical Center, Kansas City, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Medical Center, Portland, Maine
  - MedStar Washington Hospital Center, Hyattsville, Maryland
  - Union Memorial Hospital, Hyattsville, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - St. Elizabeth's Medical Center of Boston, Brighton, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Bay Regional Medical Center, Bay City, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Harper University Hospital, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St. John Hospital & Medical Center, Detroit, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. Joseph Mercy Hospital, Ypsilanti, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - North Memorial Medical Center, Robbinsdale, Minnesota
  - North Mississippi Medical Center Cardiology Associates Research, LLC, Tupelo, Mississippi
  - Boone Hospital Center, Columbia, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - St. Anthony's Medical Center, St Louis, Missouri
  - St. Patrick Hospital, Missoula, Montana
  - Nebraska Heart Hospital, Lincoln, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Cooper University Hospital, Haddon Heights, New Jersey
  - Our Lady of Lourdes Medical Center, Haddon Heights, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - St. Joseph's Regional Medical Center, Paterson, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Presbyterian Hospital, Albuquerque, New Mexico
  - St. Joseph's Hospital Health Center, Liverpool, New York
  - Long Island Jewish Medical Center, Manhasset, New York
  - Winthrop University Hospital, Mineola, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - New York Presbyterian Hospital-Cornell University, New York, New York
  - Lennox Hill Hospital,, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Strong Memorial Hospital, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Hospital, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Rex Hospital, Raleigh, North Carolina
  - WakeMed, Raleigh, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Aultman Hospital, Canton, Ohio
  - University Hospital, Cincinnati, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Tri-Health Good Samaritan Hospital, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - EMH Healthcare, Elyria, Ohio
  - Cleveland Cln Fairview Hospital, Fairview Park, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Mercy St. Vincent's Medical Center, Toledo, Ohio
  - Genesis-Good Samaritan Hospital, Zanesville, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Hillcrest Medical Center, Tulsa, Oklahoma
  - Providence St. Vincent Medical Center, Portland, Oregon
  - PeaceHealth Sacred Heart Medical Center, Springfield, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Holy Spirit Hospital, Camp Hill, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - UPMC Hamot, Erie, Pennsylvania
  - St. Mary Medical Center, Langhorne, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - UPMC Shadyside Hospital, Pittsburgh, Pennsylvania
  - Pinnacle Health at Harrisburg Hospital, Wormleysburg, Pennsylvania
  - St. Joseph Medical Center, Wyomissing, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - AnMed Health, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Sisters of Charity Providence Hospital, Columbia, South Carolina
  - Greenville Memorial Hospital of the Greenville Health System, Greenville, South Carolina
  - St. Francis Health System, Greenville, South Carolina
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Turkey Creek Medical Center, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Northwest Texas Healthcare System, Amarillo, Texas
  - Seton Medical Center Austin, Austin, Texas
  - Baylor Jack and Jane Hamilton Heart and Vascular Hospital, Dallas, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Methodist Texsan Hospital, San Antonio, Texas
  - East Texas Medical Center, Tyler, Texas
  - Trinity Mother Frances Hospital Regional Healthcare Center, Tyler, Texas
  - InterMountain Medical Center, Murray, Utah
  - Fletcher Allen Health Care, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Mary Washington Hospital, Fredericksburg, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Winchester Medical Center, Winchester, Virginia
  - St. Joseph Hospital, Bellingham, Washington
  - Providence Regional Medical Center Everett, Everett, Washington
  - Swedish Medical Center, Seattle, Washington
  - St. Mary's Medical Center, Huntington, West Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Australia (2):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria

REFERENCES:
- [Derived] Nishi T, Okada K, Kitahara H, Kameda R, Ikutomi M, Imura S, Hollak MB, Yock PG, Popma JJ, Kusano H, Cheong WF, Sudhir K, Fitzgerald PJ, Ellis SG, Kereiakes DJ, Stone GW, Honda Y, Kimura T; ABSORB III and ABSORB Japan Investigators. Intravascular ultrasound predictors of long-term outcomes following ABSORB bioresorbable scaffold implantation: A pooled analysis of the ABSORB III and ABSORB Japan trials. J Cardiol. 2021 Sep;78(3):224-229. doi: 10.1016/j.jjcc.2021.03.005. Epub 2021 Apr 21. PMID 33893022
- [Derived] Stone GW, Kimura T, Gao R, Kereiakes DJ, Ellis SG, Onuma Y, Chevalier B, Simonton C, Dressler O, Crowley A, Ali ZA, Serruys PW. Time-Varying Outcomes With the Absorb Bioresorbable Vascular Scaffold During 5-Year Follow-up: A Systematic Meta-analysis and Individual Patient Data Pooled Study. JAMA Cardiol. 2019 Dec 1;4(12):1261-1269. doi: 10.1001/jamacardio.2019.4101. PMID 31561250
- [Derived] Kereiakes DJ, Ellis SG, Metzger DC, Caputo RP, Rizik DG, Teirstein PS, Litt MR, Kini A, Kabour A, Marx SO, Popma JJ, Tan SH, Ediebah DE, Simonton C, Stone GW; ABSORB III Investigators. Clinical Outcomes Before and After Complete Everolimus-Eluting Bioresorbable Scaffold Resorption: Five-Year Follow-Up From the ABSORB III Trial. Circulation. 2019 Dec 3;140(23):1895-1903. doi: 10.1161/CIRCULATIONAHA.119.042584. Epub 2019 Sep 25. PMID 31553222
- [Derived] Kereiakes DJ, Ellis SG, Metzger C, Caputo RP, Rizik DG, Teirstein PS, Litt MR, Kini A, Kabour A, Marx SO, Popma JJ, McGreevy R, Zhang Z, Simonton C, Stone GW; ABSORB III Investigators. 3-Year Clinical Outcomes With Everolimus-Eluting Bioresorbable Coronary Scaffolds: The ABSORB III Trial. J Am Coll Cardiol. 2017 Dec 12;70(23):2852-2862. doi: 10.1016/j.jacc.2017.10.010. Epub 2017 Oct 31. PMID 29100702
- [Derived] Ali ZA, Gao R, Kimura T, Onuma Y, Kereiakes DJ, Ellis SG, Chevalier B, Vu MT, Zhang Z, Simonton CA, Serruys PW, Stone GW. Three-Year Outcomes With the Absorb Bioresorbable Scaffold: Individual-Patient-Data Meta-Analysis From the ABSORB Randomized Trials. Circulation. 2018 Jan 30;137(5):464-479. doi: 10.1161/CIRCULATIONAHA.117.031843. Epub 2017 Oct 31. PMID 29089314
- [Derived] Baron SJ, Lei Y, Chinnakondepalli K, Vilain K, Magnuson EA, Kereiakes DJ, Ellis SG, Stone GW, Cohen DJ; ABSORB III Investigators. Economic Outcomes of Bioresorbable Vascular Scaffolds Versus Everolimus-Eluting Stents in Patients Undergoing Percutaneous Coronary Intervention: 1-Year Results From the ABSORB III Trial. JACC Cardiovasc Interv. 2017 Apr 24;10(8):774-782. doi: 10.1016/j.jcin.2017.01.022. PMID 28427593
- [Derived] Stone GW, Gao R, Kimura T, Kereiakes DJ, Ellis SG, Onuma Y, Cheong WF, Jones-McMeans J, Su X, Zhang Z, Serruys PW. 1-year outcomes with the Absorb bioresorbable scaffold in patients with coronary artery disease: a patient-level, pooled meta-analysis. Lancet. 2016 Mar 26;387(10025):1277-89. doi: 10.1016/S0140-6736(15)01039-9. Epub 2016 Jan 27. PMID 26825231
- [Derived] Ellis SG, Kereiakes DJ, Metzger DC, Caputo RP, Rizik DG, Teirstein PS, Litt MR, Kini A, Kabour A, Marx SO, Popma JJ, McGreevy R, Zhang Z, Simonton C, Stone GW; ABSORB III Investigators. Everolimus-Eluting Bioresorbable Scaffolds for Coronary Artery Disease. N Engl J Med. 2015 Nov 12;373(20):1905-15. doi: 10.1056/NEJMoa1509038. Epub 2015 Oct 12. PMID 26457558
- [Derived] Kereiakes DJ, Ellis SG, Popma JJ, Fitzgerald PJ, Samady H, Jones-McMeans J, Zhang Z, Cheong WF, Su X, Ben-Yehuda O, Stone GW. Evaluation of a fully bioresorbable vascular scaffold in patients with coronary artery disease: design of and rationale for the ABSORB III randomized trial. Am Heart J. 2015 Oct;170(4):641-651.e3. doi: 10.1016/j.ahj.2015.07.013. Epub 2015 Jul 26. PMID 26386787

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first Lead-In subject (Lead-In Group ) was registered on Dec 28, 2012. A total of 2008 patients (Primary Analysis Group) were randomized into Absorb BVS arm (n = 1322) and Xience arm (n = 686) at 193 study sites between March 22, 2013 & April 3,2014 and the last 5 year follow-up visit was on May 31, 2019.
Pre-assignment Details: Of total 13,789 eligible population,11,781 patients were excluded due to,
  1. Not meeting general eligibility criteria only (n=567);
  2. Not meeting angiographic eligibility criteria only (n=10,690);
  3. Not meeting both 1 and 2 (n=64);
  4. Other reasons (n=460).
Groups:
- Absorb BVS: Subjects receiving Absorb BVS
  Absorb BVS: • Scaffold diameters: 2.5, 3.0 and 3.5 mm
  * Scaffold lengths: 8, 12, 18, and 28 mm The 3.0 x 18 mm Absorb BVS will be used for the Lead-In. Both the 8 mm and 12 mm lengths will be available for the 2.5/3.0 mm diameter Absorb BVS. Only the 12 mm length will be available for the 3.5 mm diameter.
  * The commercially approved CE marked device will be used in geographies where it is commercially available. The commercially approved CE marked 23mm Absorb BVS device will not be used in this study.
  Bioabsorbable drug eluting stent implantation for improving coronary luminal diameter in patients, including those with diabetes mellitus, with ischemic heart disease due to de novo native coronary artery lesions (length ≤ 24 mm) with a reference vessel diameter of ≥ 2.5 mm and ≤ 3.75 mm.
- XIENCE: Subjects receiving XIENCE V, XIENCE PRIME, or XIENCE Xpedition
  XIENCE: Commercially approved XIENCE Family Stent System, inclusive of XIENCE V, XIENCE PRIME, XIENCE Xpedition, XIENCE Alpine, XIENCE Pro (OUS only), and XIENCE ProX (OUS only).
  * Stent diameters: 2.5, 2.75, 3.0, 3.25, 3.5 and 4.0 mm
  * Stent lengths: 8, 12, 15, 18, 23, and 28 mm. The 3.25 mm is only available for XIENCE Xpedition
  * For geographies where these devices are commercially available, the investigational sties may use only their locally approved devices
  To improve coronary luminal diameter in patients, including those with diabetes mellitus, with ischemic heart disease due to de novo native coronary artery lesions (length ≤ 24 mm) with a reference vessel diameter of ≥ 2.5 mm and ≤ 3.75 mm.
Period: Overall Study
Arm/Group | Absorb BVS | XIENCE
Started | 1322 | 686
Completed | 1059 | 555
Not Completed | 263 | 131
Not completed — Lost to Follow-up | 151 | 68
Not completed — Withdrawal by Subject | 22 | 18
Not completed — Physician Decision | 5 | 2
Not completed — Death | 84 | 43
Not completed — Denied on premises for follow-up by law | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Absorb BVS | XIENCE | Total
Number analyzed (Participants) | 1322 | 686 | 2008
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (10.6) | 63.6 (10.3) | 63.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 388 | 205 | 593
  Male | 934 | 481 | 1415
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 23 | 73
  Not Hispanic or Latino | 1250 | 652 | 1902
  Unknown or not reported | 22 | 11 | 33
  American Indian or Alaska Native | 8 | 2 | 10
  Asian | 20 | 13 | 33
  Native Hawaiian or Other Pacific Islander | 8 | 1 | 9
  Black or African American | 70 | 34 | 104
  White | 1152 | 606 | 1758
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1318 | 683 | 2001
  Australia | 4 | 3 | 7
Hypertension Requiring Medication [Count of Participants; unit: Participants] | 1071 | 553 | 1624
Dyslipidemia Requiring Medication [Count of Participants; unit: Participants] | 1009 | 533 | 1542
Prior Coronary Intervention [Count of Participants; unit: Participants] — Population: The number of participants analyzed includes subjects who were available at that time of analysis
  Participants
    number analyzed (Participants) | 1322 | 684 | 2006
    (all) | 512 | 260 | 772
Stable Angina [Count of Participants; unit: Participants] — Population: The number of participants analyzed includes subjects who were available at that time of analysis
  Participants
    number analyzed (Participants) | 1321 | 686 | 2007
    (all) | 757 | 417 | 1174

OUTCOME MEASURES:

1. Primary Outcome: Number of Cardiac Death/TV-MI/ID-TLR (TLF)
Description: TLF is defined as composite of Cardiac Death, Myocardial Infarction (per protocol-defined MI definition), attributable to Target Vessel (TV-MI), or Ischemic-Driven Target Lesion Revascularization (ID-TLR).
Time Frame: 1 year
Population: Intent-To-Treat Population set (ITT). The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1313 | 677
Participants | 102 | 41

2. Secondary Outcome: Number of Participants With Powered Secondary Endpoint: Angina
Description: Angina is defined as the first adverse event resulting in the site diagnosis of angina.
Time Frame: 1 year
Population: The analysis will exclude angina following the index procedure through discharge, not to exceed a period of 7 days. ITT population. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1303 | 678
Participants | 238 | 125
Statistical Analysis 1: Comparison: Absorb BVS vs XIENCE; Test type: Superiority; p = 0.9256, Chi-squared

3. Secondary Outcome: Number of Participants With Powered Secondary Endpoint: All Revascularization
Description: This powered secondary endpoint is intended to assess all revascularization at 1 year and test for superiority of Absorb BVS to XIENCE. All revascularizations are comprised of TLR, TVR excluding TLR, and non-TVR.
Time Frame: 1 year
Population: ITT population. Analysis population excludes subjects who are truly lost-to-follow-up, defined as subjects who are terminated through 1 year without any DMR event (all death, all MI (regardless of MI definition), all revascularization, respectively).
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1313 | 677
Participants | 120 | 55
Statistical Analysis 1: Comparison: Absorb BVS vs XIENCE; Test type: Superiority; p = 0.5040, Fisher Exact

4. Secondary Outcome: Number of Participants With Powered Secondary Endpoint: Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: This powered secondary endpoint is intended to assess all ID-TVR at 1 year and test for superiority of Absorb BVS to XIENCE.
Time Frame: 1 year
Population: For ID-TVR, Fisher's exact test is used for superiority testing based on the ITT population. This analysis will include ~2000 subjects. ITT population. The number of participants analyzed includes subjects who had available follow up data at that time frame
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1313 | 677
Participants | 66 | 25
Statistical Analysis 1: Comparison: Absorb BVS vs XIENCE; Test type: Superiority; p = 0.2126, Fisher Exact

5. Secondary Outcome: Acute Success- Device Success (Lesion Level Analysis)
Description: Successful delivery and deployment of the study scaffold/stent at the intended target lesion and successful withdrawal of the delivery system with attainment of final in-scaffold/stent residual stenosis of less than 30% by quantitative coronary angiography (QCA) (by visual estimation if QCA unavailable). When bailout scaffold/stent is used, the success or failure of the bailout scaffold/stent delivery and deployment is not one of the criteria for device success.
Time Frame: On day 0 (the day of procedure)
Population: as for outcome 1
Measure: Number; unit: Percentage of lesions
Units Other Than Participants: Target Lesions
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1311 | 678
Number analyzed (Target Lesions) | 1355 | 704
Percentage of lesions | 94.3 | 99.3

6. Secondary Outcome: Acute Success: Procedural Success (Subject Level Analysis)
Description: Achievement of final in-scaffold/stent residual stenosis of less than 30% by QCA (by visual estimation if QCA unavailable) with successful delivery and deployment of at least one study scaffold/stent at the intended target lesion and successful withdrawal of the delivery system for all target lesions without the occurrence of cardiac death, target vessel MI or repeat TLR during the hospital stay (maximum of 7 days).
Time Frame: On day 0 (the day of procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1311 | 678
Participants | 1240 | 652

7. Secondary Outcome: Number of Death (Cardiac, Vascular, Non-cardiovascular)
Description: DEATH (Per ARC Circulation) : All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Specifically, any unexpected death even in patients with coexisting potentially fatal non-cardiac disease (e.g. cancer, infection) should be classified as cardiac.
  Cardiac death (CD): Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
Time Frame: 0 to 5 years
Population: ITT set. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1187 | 612
Participants | 85 | 44

8. Secondary Outcome: Number of Participants With All Myocardial Infarction (MI)
Description: * Attributable to target vessel (TV-MI)
  * Not attributable to target vessel (NTV-MI)
Time Frame: 0 to 5 years
Population: ITT set. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1187 | 612
Participants | 159 | 69

9. Secondary Outcome: Number of Participants With All Target Lesion Revascularization (TLR)
Description: TLR is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. All TLR should be classified prospectively as ischemia driven (ID-TLR) or not ischemia driven (NID-TLR) by the investigator prior to repeat angiography.
  The target lesion is defined as the treated segment from 5 mm proximal to the stent and to 5 mm distal to the stent.
Time Frame: 0 to 5 years
Population: ITT set. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1187 | 612
Participants | 118 | 51

10. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR) Excluding Target Lesion Revascularization (TLR)
Description: TVR is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion which includes upstream and downstream branches and the target lesion itself.
Time Frame: 0 to 5 years
Population: ITT set. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1187 | 612
Participants | 108 | 40

11. Secondary Outcome: Number of Participants With All Revascularization
Description: All revascularization endpoint is comprised of TLR, TVR excluding TLR, and non-TVR.
Time Frame: 0 to 5 years
Population: ITT set. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1187 | 612
Participants | 255 | 114

12. Secondary Outcome: Number of Death/All MI
Description: All deaths includes Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
  Myocardial Infarction (MI) - Q wave MI: Development of new, pathological Q wave on the ECG.
  -Non-Q wave MI: Those MIs which are not Q-wave MI
Time Frame: 0 to 5 years
Population: ITT set. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1187 | 612
Participants | 230 | 101

13. Secondary Outcome: Number of Cardiac Death/All MI
Description: as for outcome 12
Time Frame: 0 to 5 years
Population: ITT set. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1187 | 612
Participants | 185 | 81

14. Secondary Outcome: Number of Cardiac Death/TV-MI/ID-TLR (TLF)
Description: Target Lesion Failure is composite of Cardiac death/ Target Vessel Myocardial Infarction (TV-MI)/ Ischemic-Driven Target Lesion Revascularization (ID-TLR).
Time Frame: 0 to 5 years
Population: ITT set. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1187 | 612
Participants | 220 | 98

15. Secondary Outcome: Number of Cardiac Death/All MI/ID-TLR (Major Adverse Cardiac Events-MACE)
Description: Major adverse cardiac events (MACE) is defined as the composite of cardiac death, all myocardial infarction, and ischemic driven target lesion revascularization (ID-TLR).
Time Frame: 0 to 5 years
Population: ITT set. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1187 | 612
Participants | 245 | 113

16. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: Target Vessel Failure (TVF) is the composite of Cardiac Death, Myocardial infarction (MI) or Ischemic-Driven Target Vessel Revascularization (ID-TVR).
Time Frame: 0 to 5 years
Population: ITT set. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1187 | 612
Participants | 290 | 128

17. Secondary Outcome: Number of Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization.
Time Frame: 0 to 5 years
Population: ITT set. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1187 | 612
Participants | 378 | 168

18. Secondary Outcome: Number of Participants With Acute Stent/Scaffold Thrombosis (Per ARC Definition)
Description: Stent Thrombosis should be reported as a cumulative value at the different time points and with the different separate time points. Time 0 is defined as the time point after the guiding catheter has been removed and the subject left the Catheterization lab.
  Timing :
  Acute : 0 - 24 hours post stent implantation; Subacute : >24 hours - 30 days post stent implantation; Late : 30 days - 1 year post stent implantation; Very late : >1 year post stent implantation.
  Evidence:
  Definite stent thrombosis is considered to have occurred by either angiographic or pathologic confirmation.
  Probable stent thrombosis is considered to have occurred after intracoronary stenting in case of Any unexplained death within the first 30 days or Irrespective of the time after the index procedure, any MI that is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause.
Time Frame: ≤ 1 Day
Population: Analyzed population excludes subjects who are truly lost-to-follow-up, defined as subjects who are terminated through a given time point without any Stent/Scaffold Thrombosis event. ITT population. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1319 | 686
Participants
  Definite/Probable | 3 | 4
  Definite | 3 | 4
  Probable | 0 | 0

19. Secondary Outcome: Number of Participants With Acute/Subacute Stent/Scaffold Thrombosis (Per ARC Definition)
Description: as for outcome 18
Time Frame: 0 to 30 Days
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1314 | 686
Participants
  Definite/Probable | 14 | 5
  Definite | 12 | 5
  Probable | 2 | 0

20. Secondary Outcome: Number of Participants With Subacute Stent/Scaffold Thrombosis
Description: as for outcome 18
Time Frame: >1 to 30 Days
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1314 | 686
Participants
  Definite/Probable | 12 | 1
  Definite | 10 | 1
  Probable | 2 | 0

21. Secondary Outcome: Number of Participants With Late Stent/Scaffold Thrombosis (Per ARC Definition)
Description: Stent Thrombosis should be reported as a cumulative value at the different time points and with the different separate time points. Time 0 is defined as the time point after the guiding catheter has been removed and the subject left the Catheterization lab.
  Timing :
  Acute : 0 - 24 hours post stent implantation; Subacute : >24 hours - 30 days post stent implantation; Late : 30 days - 1 year post stent implantation; Very late : >1 year post stent implantation.
  Evidence:
  Definite stent thrombosis is considered to have occurred by either angiographic or pathologic confirmation.
  Probable stent thrombosis is considered to have occurred after intracoronary stenting in case of
  * Any unexplained death within the first 30 days or
  * Irrespective of the time after the index procedure, any MI that is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause.
Time Frame: 31 to 365 Days
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1289 | 672
Participants
  Definite/Probable | 6 | 0
  Definite | 6 | 0
  Probable | 0 | 0

22. Secondary Outcome: Number of Participants With Very Late Stent /Scaffold Thrombosis (Per ARC Definition)
Description: as for outcome 21
Time Frame: 366 to 393 Days
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1289 | 672
Participants
  Definite/Probable | 0 | 0
  Definite | 0 | 0
  Probable | 0 | 0

23. Secondary Outcome: Number of Participants With Cumulative Stent/Scaffold Thrombosis
Description: as for outcome 21
Time Frame: 0 to 1853 Days
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1072 | 558
Participants
  Definite/Probable | 32 | 7
  Definite | 30 | 7
  Probable | 2 | 0

24. Secondary Outcome: Pre-Procedure Minimum Lumen Diameter (MLD)
Description: Angiographic endpoint Minimum lumen diameter is defined as the shortest diameter through the center point of the lumen.
Time Frame: < or = 1 day
Population: ITT population. The number of participants analyzed includes subjects who had available follow-up data at that time frame. The analysis excludes subjects who are truly lost to follow-up.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target Lesions
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1322 | 686
Number analyzed (Target Lesions) | 1380 | 708
Millimeter | 0.92 (0.37) | 0.90 (0.34)

25. Secondary Outcome: Pre-Procedure Percent Diameter Stenosis (%DS)
Description: Percent Diameter Stenosis is defined as the value calculated as 100 * (1 - Minimum Luminal Diameter (MLD)/Reference vessel diameter (RVD)) using the mean values from two orthogonal views (when possible) by quantitative coronary angiography (QCA).
Time Frame: < or = 1 day
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Percent Diameter stenosis
Units Other Than Participants: Target Lesions
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1322 | 686
Number analyzed (Target Lesions) | 1380 | 708
Percent Diameter stenosis | 65.25 (12.48) | 65.90 (11.66)

26. Secondary Outcome: Post-Procedure In-Segment Minimum Lumen Diameter (MLD)
Description: Angiographic endpoint. Minimum lumen diameter is defined as the shortest diameter through the center point of the lumen.
  In- Segment is defined as, within the margins of the stent or scaffold and 5 mm proximal and 5 mm distal to the stent or scaffold.
Time Frame: ≤ 7 days post index procedure
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target Lesions
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1322 | 686
Number analyzed (Target Lesions) | 1374 | 706
Millimeter | 2.15 (0.41) | 2.14 (0.43)

27. Secondary Outcome: Post-Procedure In-Segment Percent Diameter Stenosis (%DS)
Description: Angiographic endpoint. Percent Diameter Stenosis is defined as the value calculated as 100 * (1 - Minimum Luminal Diameter (MLD)/Reference vessel diameter (RVD)) using the mean values from two orthogonal views (when possible) by quantitative coronary angiography (QCA).
  In- Segment is defined as, within the margins of the stent or scaffold and 5 mm proximal and 5 mm distal to the stent or scaffold.
Time Frame: ≤ 7 days post index procedure
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Percent Diameter stenosis
Units Other Than Participants: Target Lesions
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1322 | 686
Number analyzed (Target Lesions) | 1374 | 706
Percent Diameter stenosis | 20.04 (7.94) | 19.82 (8.20)

28. Secondary Outcome: Post-Procedure In-Device Minimum Lumen Diameter (MLD)
Description: as for outcome 26
Time Frame: ≤ 7 days post index procedure
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target Lesions
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1322 | 686
Number analyzed (Target Lesions) | 1373 | 706
Millimeter | 2.37 (0.40) | 2.49 (0.40)

29. Secondary Outcome: Post-Procedure In-Device Percent Diameter Stenosis (%DS)
Description: Angiographic endpoint. Percent Diameter Stenosis is defined as the value calculated as 100 * (1 - Minimum Luminal Diameter (MLD)/Reference vessel diameter (RVD)) using the mean values from two orthogonal views (when possible) by quantitative coronary angiography (QCA).
Time Frame: ≤ 7 days post index procedure
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Percent Diameter stenosis
Units Other Than Participants: Target Lesions
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1322 | 686
Number analyzed (Target Lesions) | 1369 | 702
Percent Diameter stenosis | 11.62 (8.77) | 6.41 (8.91)

30. Secondary Outcome: Post-Procedure In-Device Acute Gain
Description: The acute gain was defined as the difference between post- and pre procedural minimal lumen diameter (MLD).
Time Frame: ≤ 7 days post index procedure
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Target Lesions
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1322 | 686
Number analyzed (Target Lesions) | 1372 | 706
mm | 1.45 (0.45) | 1.59 (0.44)

31. Secondary Outcome: Powered Imaging Cohort Secondary Endpoint: The Instent/Scaffold Mean Lumen Area Change, From Post Procedure to 3 Years by Intravascular Ultrasound (IVUS)
Description: * Mean lumen area measured after nitrate infusions, superiority test, ~300 pooled subjects.
  * Pooled IVUS subjects (~300 subjects): 150 subjects from the Imaging Cohort of ABSORB III RCT and 150 subjects from ABSORB Japan RCT.
Time Frame: From Post procedure to 3 Years
Population: The full analysis set (FAS) population is defined as the patients wherein the target lesion was treated with the assigned device.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Lesions
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 188 | 93
Number analyzed (Lesions) | 119 | 65
mm^2 | -0.30 (1.32) | -0.60 (0.91)
Statistical Analysis 1: Comparison: Absorb BVS vs XIENCE; Test type: Superiority; p = 0.0665, Chi-squared

32. Secondary Outcome: Optical Coherence Tomography (OCT) Endpoint: Mean Neointimal Area (NIA)
Description: All OCT endpoints will be collected for within the device and within the treated segment: Descriptive analysis of strut, lesion and vessel morphology Mean neointimal area (NIA) - Apposed to the vessel wall with neointimal coverage Apposed to vessel wall without neointimal coverage Incomplete apposition to vessel wall with neointimal coverage Incomplete apposition to vessel wall without neointimal coverage Lumen area/volume stenosis % Mean/minimal device area Mean/minimal luminal area/volume Mean strut area/volume Persisting incomplete apposition, late incomplete apposition at 3 years (if analyzable) OCT analysis for subjects with jailed side branch Descriptive analyses from 3-dimensional OCT reconstructions
Time Frame: 3 Years
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Leisions
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 33 | 16
Number analyzed (Leisions) | 21 | 10
mm^2 | 1.12 (0.48) | 1.19 (0.61)

33. Secondary Outcome: Optical Coherence Tomography (OCT) Endpoint: Mean Device Area, Adluminal
Description: as for outcome 32
Time Frame: 3 Years
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Leisions
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 33 | 16
Number analyzed (Leisions) | 33 | 16
mm^2
  Post-procedure: number analyzed (Leisions) | 26 | 14
  Post-procedure | 6.89 (1.98) | 7.25 (1.51)
  3 Years: number analyzed (Leisions) | 21 | 10
  3 Years | 7.70 (2.54) | 7.24 (1.90)

34. Secondary Outcome: Optical Coherence Tomography (OCT) Endpoint: Mean Lumen Area
Description: as for outcome 32
Time Frame: 3 Years
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Leisions
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 33 | 16
Number analyzed (Leisions) | 33 | 16
mm^2
  Post-procedure: number analyzed (Leisions) | 26 | 14
  Post-procedure | 7.99 (2.12) | 7.50 (1.46)
  3 Years: number analyzed (Leisions) | 21 | 10
  3 Years | 6.67 (2.36) | 6.06 (1.73)

35. Secondary Outcome: Optical Coherence Tomography (OCT) Endpoint: Minimal Lumen Area
Description: as for outcome 32
Time Frame: 3 Years
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Leisions
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 33 | 16
Number analyzed (Leisions) | 33 | 16
mm^2
  Post-procedure: number analyzed (Leisions) | 26 | 14
  Post-procedure | 6.47 (1.82) | 6.07 (1.46)
  3 Years: number analyzed (Leisions) | 21 | 10
  3 Years | 4.95 (1.78) | 4.54 (1.40)

36. Secondary Outcome: Optical Coherence Tomography (OCT) Endpoint: Percentage of Malapposition Struts
Description: as for outcome 32
Time Frame: 3 Years
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Percentage of Malapposition Struts
Units Other Than Participants: Leisions
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 33 | 16
Number analyzed (Leisions) | 33 | 16
Percentage of Malapposition Struts
  Post-procedure: number analyzed (Leisions) | 26 | 14
  Post-procedure | 7.42 (5.49) | 7.64 (6.26)
  3 Years: number analyzed (Leisions) | 21 | 10
  3 Years | 0.32 (0.99) | 0.07 (0.22)

37. Other Pre Specified Outcome: Patient Reported Outcomes (PRO): Overall Health Status
Description: Overall health status assessed using the EuroQoL 5D (EQ-5D™).
  EQ-5D:
  * Scale range: 0 to 1
  * Higher values represent better outcomes
  * Health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Subscale scores are summed to obtain total/overall health status.
  A scoring algorithm was used to combine the sub-scores from each of the 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), and generate a single index ranging from 0 to 1
Time Frame: Baseline
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1249 | 651
score on a scale | 0.77 (0.2) | 0.77 (0.20)

38. Other Pre Specified Outcome: Patient Reported Outcomes (PRO): Overall Health Status
Description: as for outcome 37
Time Frame: 1 month
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1231 | 647
score on a scale | 0.85 (0.18) | 0.85 (0.18)

39. Other Pre Specified Outcome: Patient Reported Outcomes (PRO): Overall Health Status
Description: as for outcome 37
Time Frame: 12 months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1087 | 567
score on a scale | 0.83 (0.20) | 0.83 (0.19)

40. Other Pre Specified Outcome: Patient Reported Outcomes (PRO): Anxiety
Description: Anxiety assessed using the Generalized Anxiety Disorder scale (GAD-7).
  GAD-7:
  * Scale range: 0 to 21
  * Lower values represent better outcomes
  * No subscales
Time Frame: Baseline
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1009 | 530
score on a scale | 5.92 (5.86) | 6.34 (6.07)

41. Other Pre Specified Outcome: Patient Reported Outcomes (PRO): Anxiety
Description: as for outcome 40
Time Frame: 1 month
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1067 | 556
score on a scale | 3.39 (4.64) | 3.33 (4.61)

42. Other Pre Specified Outcome: Patient Reported Outcomes (PRO): Anxiety
Description: as for outcome 40
Time Frame: 12 months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 911 | 482
score on a scale | 3.92 (4.99) | 4.04 (5.08)

43. Other Pre Specified Outcome: Patient Reported Outcomes (PRO): Disease-Specific Quality of Life
Description: Disease-Specific quality of life assessed using the Seattle Angina Questionnaire (SAQ)
  Seattle Angina Questionnaire (SAQ): Each scale is transformed to a score of 0 to 100, where higher scores indicate better function (eg, less physical limitation, less angina, and better quality of life).
Time Frame: Baseline
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1195 | 617
score on a scale | 67.67 (20.20) | 67.11 (19.17)

44. Other Pre Specified Outcome: Patient Reported Outcomes (PRO): Disease-Specific Quality of Life
Description: Disease-Specific quality of life in hospital baseline and at 1 year assessed using the Seattle Angina Questionnaire (SAQ).
  Seattle Angina Questionnaire (SAQ): Each scale is transformed to a score of 0 to 100, where higher scores indicate better function (eg, less physical limitation, less angina, and better quality of life).
Time Frame: 1 month
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1131 | 589
score on a scale | 87.10 (14.27) | 86.98 (14.16)

45. Other Pre Specified Outcome: Patient Reported Outcomes (PRO): Disease-Specific Quality of Life
Description: as for outcome 44
Time Frame: 12 months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1014 | 514
score on a scale | 87.05 (13.91) | 86.42 (14.45)

46. Other Pre Specified Outcome: Patient Reported Outcomes (PRO): Dyspnea Severity
Description: Dyspnea severity assessed using the Rose Dyspnea Scale (RDS).
  Rose Dyspnea Scale:
  * Scale range: 0 to 4
  * Lower values represent better outcomes (higher scores indicate worse dyspnea)
  * No subscales
Time Frame: Baseline
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1242 | 651
score on a scale | 1.66 (1.48) | 1.65 (1.46)

47. Other Pre Specified Outcome: Patient Reported Outcomes (PRO): Dyspnea Severity
Description: as for outcome 46
Time Frame: 1 month
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1220 | 636
score on a scale | 0.81 (1.24) | 0.88 (1.29)

48. Other Pre Specified Outcome: Patient Reported Outcomes (PRO): Dyspnea Severity
Description: as for outcome 46
Time Frame: 12 months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1080 | 568
score on a scale | 0.94 (1.26) | 0.99 (1.30)

49. Other Pre Specified Outcome: Landmark Analysis on TLF and Components
Description: TLF is defined as composite of Cardiac Death, Myocardial Infarction (per protocol-defined MI definition), attributable to Target Vessel (TVMI), or Ischemic-Driven Target Lesion Revascularization (ID-TLR).
Time Frame: 3-4 years
Population: ITT set. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1202 | 610
Participants | 38 | 16

50. Other Pre Specified Outcome: Landmark Analysis on TLF and Components
Description: as for outcome 49
Time Frame: 3-5 years
Population: ITT set. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1108 | 580
Participants | 60 | 38

51. Other Pre Specified Outcome: Landmark Analysis on Cumulative Scaffold Thrombosis/Stent Thrombosis (Per ARC Definition, Definite and Probable)
Description: as for outcome 21
Time Frame: 3-4 years
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1180 | 607
Participants
  Definite/Probable | 1 | 1
  Definite | 1 | 1
  Probable | 0 | 0

52. Other Pre Specified Outcome: Landmark Analysis on Cumulative Scaffold Thrombosis/Stent Thrombosis (Per ARC Definition, Definite and Probable)
Description: as for outcome 21
Time Frame: 3-5 years
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE
Number analyzed (Participants) | 1059 | 556
Participants
  Definite/Probable | 1 | 2
  Definite | 1 | 2
  Probable | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Absorb BVS | XIENCE
All-Cause Mortality (participants affected / at risk) | 85/1322 | 44/686
Serious Adverse Events (participants affected / at risk) | 801/1322 | 398/686
Other Adverse Events (participants affected / at risk) | 1174/1322 | 601/686
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Absorb BVS (N=1322) | XIENCE (N=686)
ANAEMIA (Blood and lymphatic system disorders) | 7 | 7
ANAEMIA OF CHRONIC DISEASE (Blood and lymphatic system disorders) | 0 | 1
COAGULOPATHY (Blood and lymphatic system disorders) | 0 | 2
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 2 | 3
HEPARIN-INDUCED THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0
IRON DEFICIENCY ANEMIA (Blood and lymphatic system disorders) | 1 | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 2 | 1
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 2 | 0
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
NORMOCHROMIC NORMOCYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 6 | 5
ACUTE LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 49 | 21
ANGINA PECTORIS (Cardiac disorders) | 161 | 87
ANGINA UNSTABLE (Cardiac disorders) | 68 | 28
AORTIC VALVE DISEASE (Cardiac disorders) | 2 | 0
AORTIC VALVE STENOSIS (Cardiac disorders) | 6 | 2
ARRHYTHMIA (Cardiac disorders) | 1 | 2
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 2 | 0
ARTERIOSPASM CORONARY (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 52 | 21
ATRIAL FLUTTER (Cardiac disorders) | 6 | 2
ATRIAL TACHYCARDIA (Cardiac disorders) | 0 | 1
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 3 | 0
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 | 1
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 4 | 0
BRADYCARDIA (Cardiac disorders) | 9 | 2
BUNDLE BRANCH BLOCK (Cardiac disorders) | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 10 | 6
CARDIAC FAILURE (Cardiac disorders) | 8 | 4
CARDIAC FAILURE ACUTE (Cardiac disorders) | 5 | 1
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 2 | 3
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 32 | 25
CARDIAC TAMPONADE (Cardiac disorders) | 1 | 0
CARDIAC VALVE DISEASE (Cardiac disorders) | 2 | 0
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 2 | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 1 | 3
CARDIOMYOPATHY (Cardiac disorders) | 1 | 1
CARDIORENAL SYNDROME (Cardiac disorders) | 1 | 0
CHRONIC LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1 | 0
CONDUCTION DISORDER (Cardiac disorders) | 0 | 1
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 38 | 24
CORONARY ARTERY DISSECTION (Cardiac disorders) | 22 | 12
CORONARY ARTERY EMBOLISM (Cardiac disorders) | 2 | 2
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 4 | 2
CORONARY ARTERY PERFORATION (Cardiac disorders) | 5 | 3
CORONARY ARTERY STENOSIS (Cardiac disorders) | 20 | 13
CORONARY OSTIAL STENOSIS (Cardiac disorders) | 1 | 0
DRESSLER'S SYNDROME (Cardiac disorders) | 0 | 2
IN-STENT CORONARY ARTERY RESTENOSIS (Cardiac disorders) | 4 | 5
INTRACARDIAC THROMBUS (Cardiac disorders) | 1 | 0
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 3 | 1
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 | 1
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 5 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 52 | 23
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 3 | 0
PALPITATIONS (Cardiac disorders) | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 5 | 1
PERICARDITIS (Cardiac disorders) | 1 | 1
PRINZMETAL ANGINA (Cardiac disorders) | 2 | 0
SICK SINUS SYNDROME (Cardiac disorders) | 6 | 3
SINUS ARRHYTHMIA (Cardiac disorders) | 0 | 1
SINUS BRADYCARDIA (Cardiac disorders) | 1 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 5 | 2
TACHYCARDIA (Cardiac disorders) | 1 | 1
TORSADE DE POINTES (Cardiac disorders) | 1 | 0
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 | 1
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 3 | 0
VENTRICULAR FIBRILLATION (Cardiac disorders) | 5 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 8 | 3
CYSTIC LYMPHANGIOMA (Congenital, familial and genetic disorders) | 1 | 0
PULMONARY ARTERIOVENOUS FISTULA (Congenital, familial and genetic disorders) | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 5 | 1
AMAUROSIS FUGAX (Eye disorders) | 1 | 0
CATARACT (Eye disorders) | 0 | 3
CATARACT NUCLEAR (Eye disorders) | 1 | 0
DIPLOPIA (Eye disorders) | 1 | 0
GLAUCOMA (Eye disorders) | 2 | 0
MACULAR OEDEMA (Eye disorders) | 1 | 0
PAPILLOEDEMA (Eye disorders) | 1 | 0
POSTERIOR CAPSULE OPACIFICATION (Eye disorders) | 1 | 0
RETINAL DETACHMENT (Eye disorders) | 1 | 1
RETINAL HAEMORRHAGE (Eye disorders) | 0 | 1
VISION BLURRED (Eye disorders) | 1 | 0
ABDOMINAL HERNIA (Gastrointestinal disorders) | 3 | 3
ABDOMINAL HERNIA OBSTRUCTIVE (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 3
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 3
ABDOMINAL WALL HAEMATOMA (Gastrointestinal disorders) | 1 | 0
ALCOHOLIC PANCREATITIS (Gastrointestinal disorders) | 0 | 1
COELIAC ARTERY STENOSIS (Gastrointestinal disorders) | 1 | 0
COLITIS (Gastrointestinal disorders) | 2 | 1
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 1 | 1
CONSTIPATION (Gastrointestinal disorders) | 2 | 0
CROHN'S DISEASE (Gastrointestinal disorders) | 2 | 0
DENTAL CARIES (Gastrointestinal disorders) | 1 | 0
DIABETIC GASTROPARESIS (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 3 | 2
DIVERTICULUM (Gastrointestinal disorders) | 0 | 1
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 2 | 1
DUODENAL ULCER (Gastrointestinal disorders) | 1 | 0
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 5 | 1
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 1 | 0
FAECALOMA (Gastrointestinal disorders) | 1 | 0
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 2 | 2
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 2 | 0
GASTRITIS (Gastrointestinal disorders) | 2 | 0
GASTROINTESTINAL ANGIODYSPLASIA (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 13 | 13
GASTROINTESTINAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 5 | 0
HAEMATEMESIS (Gastrointestinal disorders) | 1 | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 | 0
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 0
HIATUS HERNIA (Gastrointestinal disorders) | 1 | 1
ILEUS (Gastrointestinal disorders) | 1 | 2
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 3 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 2 | 3
INTESTINAL MASS (Gastrointestinal disorders) | 2 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 2
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 1 | 0
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 2
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 1 | 0
MELAENA (Gastrointestinal disorders) | 1 | 1
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
OESOPHAGEAL ACHALASIA (Gastrointestinal disorders) | 0 | 1
OESOPHAGITIS (Gastrointestinal disorders) | 1 | 0
PANCREATIC CYST (Gastrointestinal disorders) | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 1 | 2
PANCREATITIS ACUTE (Gastrointestinal disorders) | 2 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 2
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 3 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 | 6
SMALL INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 | 1
UMBILICAL HERNIA (Gastrointestinal disorders) | 2 | 0
UMBILICAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 1 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 3 | 4
ABASIA (General disorders) | 0 | 1
ADVERSE DRUG REACTION (General disorders) | 3 | 1
ASTHENIA (General disorders) | 5 | 0
CARDIAC DEATH (General disorders) | 1 | 0
CATHETER SITE HAEMATOMA (General disorders) | 1 | 1
CATHETER SITE HAEMORRHAGE (General disorders) | 1 | 2
CATHETER SITE PAIN (General disorders) | 0 | 2
CHEST DISCOMFORT (General disorders) | 10 | 8
CHEST PAIN (General disorders) | 40 | 18
DEATH (General disorders) | 10 | 6
DEVICE ELECTRICAL FINDING (General disorders) | 0 | 1
DEVICE FAILURE (General disorders) | 1 | 1
DEVICE MALFUNCTION (General disorders) | 1 | 0
DEVICE OCCLUSION (General disorders) | 1 | 0
DROWNING (General disorders) | 1 | 0
DRUG INTOLERANCE (General disorders) | 1 | 0
DRUG WITHDRAWAL SYNDROME (General disorders) | 1 | 0
HERNIA (General disorders) | 0 | 1
HERNIA OBSTRUCTIVE (General disorders) | 1 | 0
IMPAIRED HEALING (General disorders) | 0 | 1
MEDICAL DEVICE SITE REACTION (General disorders) | 1 | 0
MULTI-ORGAN FAILURE (General disorders) | 1 | 2
NON-CARDIAC CHEST PAIN (General disorders) | 84 | 51
OEDEMA PERIPHERAL (General disorders) | 1 | 0
PAIN (General disorders) | 1 | 0
PELVIC MASS (General disorders) | 0 | 2
PYREXIA (General disorders) | 6 | 3
SUDDEN CARDIAC DEATH (General disorders) | 0 | 1
SURGICAL FAILURE (General disorders) | 1 | 0
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 3 | 1
THROMBOSIS IN DEVICE (General disorders) | 9 | 6
BILE DUCT STONE (Hepatobiliary disorders) | 2 | 0
CHOLANGITIS (Hepatobiliary disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 3 | 2
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 2 | 4
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 7 | 3
GALLBLADDER DISORDER (Hepatobiliary disorders) | 1 | 0
HEPATIC LESION (Hepatobiliary disorders) | 2 | 1
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 1 | 0
ALLERGY TO ARTHROPOD STING (Immune system disorders) | 1 | 1
ABDOMINAL ABSCESS (Infections and infestations) | 0 | 1
ABSCESS NECK (Infections and infestations) | 1 | 0
APPENDICITIS (Infections and infestations) | 4 | 2
APPENDICITIS PERFORATED (Infections and infestations) | 1 | 0
ARTHRITIS BACTERIAL (Infections and infestations) | 1 | 0
ARTHRITIS INFECTIVE (Infections and infestations) | 1 | 0
BACTERAEMIA (Infections and infestations) | 4 | 0
BACTERIAL INFECTION (Infections and infestations) | 0 | 1
BACTERIAL SEPSIS (Infections and infestations) | 0 | 2
BREAST CELLULITIS (Infections and infestations) | 1 | 0
BRONCHITIS (Infections and infestations) | 10 | 6
BRONCHITIS VIRAL (Infections and infestations) | 1 | 0
CATHETER SITE ABSCESS (Infections and infestations) | 2 | 0
CATHETER SITE CELLULITIS (Infections and infestations) | 1 | 0
CATHETER SITE INFECTION (Infections and infestations) | 1 | 0
CELLULITIS (Infections and infestations) | 11 | 11
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 0 | 2
CLOSTRIDIAL INFECTION (Infections and infestations) | 1 | 1
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 2 | 2
CYSTITIS (Infections and infestations) | 1 | 0
DIABETIC FOOT INFECTION (Infections and infestations) | 1 | 0
DIVERTICULITIS (Infections and infestations) | 5 | 3
ENDOCARDITIS (Infections and infestations) | 1 | 0
ENTEROCOCCAL SEPSIS (Infections and infestations) | 0 | 1
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 | 0
FUNGAL INFECTION (Infections and infestations) | 0 | 1
GANGRENE (Infections and infestations) | 1 | 1
GASTROENTERITIS (Infections and infestations) | 6 | 3
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 2
GENITAL INFECTION FEMALE (Infections and infestations) | 1 | 0
HERPES ZOSTER (Infections and infestations) | 1 | 1
HIV INFECTION (Infections and infestations) | 1 | 0
IMPLANT SITE INFECTION (Infections and infestations) | 1 | 0
INFECTED DERMAL CYST (Infections and infestations) | 1 | 0
INFECTED SKIN ULCER (Infections and infestations) | 0 | 1
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 1 | 0
INFLUENZA (Infections and infestations) | 3 | 3
KIDNEY INFECTION (Infections and infestations) | 3 | 0
LOBAR PNEUMONIA (Infections and infestations) | 1 | 1
LOCALISED INFECTION (Infections and infestations) | 0 | 3
LUNG ABSCESS (Infections and infestations) | 0 | 1
MENINGITIS ASEPTIC (Infections and infestations) | 1 | 0
METAPNEUMOVIRUS INFECTION (Infections and infestations) | 1 | 0
MYCOBACTERIUM ABSCESSUS INFECTION (Infections and infestations) | 1 | 0
ORAL FUNGAL INFECTION (Infections and infestations) | 1 | 0
ORCHITIS (Infections and infestations) | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 3 | 4
PERITONITIS (Infections and infestations) | 0 | 1
PERITONSILLAR ABSCESS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 25 | 19
PNEUMONIA ADENOVIRAL (Infections and infestations) | 1 | 0
PNEUMONIA BACTERIAL (Infections and infestations) | 2 | 0
PNEUMONIA NECROTISING (Infections and infestations) | 1 | 0
PNEUMONIA PRIMARY ATYPICAL (Infections and infestations) | 1 | 0
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 1 | 0
POST PROCEDURAL CELLULITIS (Infections and infestations) | 1 | 0
POST PROCEDURAL INFECTION (Infections and infestations) | 1 | 0
POST PROCEDURAL PNEUMONIA (Infections and infestations) | 1 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 | 1
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 1 | 0
SEPSIS (Infections and infestations) | 14 | 10
SEPSIS SYNDROME (Infections and infestations) | 2 | 0
SEPTIC ENCEPHALOPATHY (Infections and infestations) | 0 | 1
SEPTIC SHOCK (Infections and infestations) | 2 | 1
SPINAL CORD INFECTION (Infections and infestations) | 1 | 0
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 2
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0
URINARY TRACT INFECTION (Infections and infestations) | 9 | 7
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 1 | 1
UROSEPSIS (Infections and infestations) | 3 | 4
VIRAL INFECTION (Infections and infestations) | 2 | 0
VIRAL LABYRINTHITIS (Infections and infestations) | 0 | 1
WOUND INFECTION (Infections and infestations) | 1 | 2
WOUND INFECTION BACTERIAL (Infections and infestations) | 0 | 1
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 0 | 1
ACETABULUM FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 2 | 2
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 3 | 2
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 3
BURNS THIRD DEGREE (Injury, poisoning and procedural complications) | 0 | 1
CARDIAC PROCEDURE COMPLICATION (Injury, poisoning and procedural complications) | 1 | 1
CEREBRAL HAEMORRHAGE TRAUMATIC (Injury, poisoning and procedural complications) | 2 | 0
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
COLON INJURY (Injury, poisoning and procedural complications) | 1 | 0
CONCUSSION (Injury, poisoning and procedural complications) | 1 | 0
CONTRAST MEDIA ALLERGY (Injury, poisoning and procedural complications) | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 2 | 0
CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 51 | 15
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 3 | 0
CYSTITIS RADIATION (Injury, poisoning and procedural complications) | 1 | 0
DEEP VEIN THROMBOSIS POSTOPERATIVE (Injury, poisoning and procedural complications) | 2 | 0
EXPOSURE TO TOXIC AGENT (Injury, poisoning and procedural complications) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 9 | 7
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 | 2
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 3 | 0
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
GASTROINTESTINAL ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 0 | 1
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 4 | 2
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 2
ILIOTIBIAL BAND SYNDROME (Injury, poisoning and procedural complications) | 0 | 1
IN-STENT ARTERIAL RESTENOSIS (Injury, poisoning and procedural complications) | 0 | 1
IN-STENT CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 7 | 5
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 3 | 0
INJURY (Injury, poisoning and procedural complications) | 1 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 | 1
LACERATION (Injury, poisoning and procedural complications) | 1 | 0
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 1 | 1
LIMB TRAUMATIC AMPUTATION (Injury, poisoning and procedural complications) | 1 | 0
MENISCUS LESION (Injury, poisoning and procedural complications) | 4 | 1
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 2 | 0
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 1 | 0
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 0 | 1
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
PLAQUE SHIFT (Injury, poisoning and procedural complications) | 1 | 3
POST CONCUSSION SYNDROME (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 2
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 2
POST PROCEDURAL MYOCARDIAL INFARCTION (Injury, poisoning and procedural complications) | 7 | 5
POST PROCEDURAL STROKE (Injury, poisoning and procedural complications) | 1 | 0
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 2 | 0
POSTOPERATIVE ADHESION (Injury, poisoning and procedural complications) | 1 | 0
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
PROCEDURAL DIZZINESS (Injury, poisoning and procedural complications) | 1 | 0
PROCEDURAL HEADACHE (Injury, poisoning and procedural complications) | 1 | 0
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 0 | 1
PROCEDURAL VOMITING (Injury, poisoning and procedural complications) | 1 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
RESPIRATORY FUME INHALATION DISORDER (Injury, poisoning and procedural complications) | 1 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 2 | 2
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 4 | 0
SEROMA (Injury, poisoning and procedural complications) | 1 | 0
SKULL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
SNAKE BITE (Injury, poisoning and procedural complications) | 1 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 4 | 2
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 6 | 3
TENDON INJURY (Injury, poisoning and procedural complications) | 0 | 1
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
THERMAL BURN (Injury, poisoning and procedural complications) | 1 | 0
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 | 2
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
TRAUMATIC HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1
ULNA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
URINARY RETENTION POSTOPERATIVE (Injury, poisoning and procedural complications) | 3 | 0
VASCULAR GRAFT OCCLUSION (Injury, poisoning and procedural complications) | 2 | 1
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 7 | 3
WOUND (Injury, poisoning and procedural complications) | 1 | 0
WOUND EVISCERATION (Injury, poisoning and procedural complications) | 1 | 0
WOUND HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
WRIST FRACTURE (Injury, poisoning and procedural complications) | 2 | 1
BIOPSY LUNG (Investigations) | 0 | 1
BLOOD CREATINE INCREASED (Investigations) | 1 | 0
BLOOD CREATINE PHOSPHOKINASE MB INCREASED (Investigations) | 2 | 0
BLOOD CREATININE INCREASED (Investigations) | 3 | 0
BLOOD PRESSURE INCREASED (Investigations) | 1 | 1
BLOOD PRESSURE SYSTOLIC INCREASED (Investigations) | 1 | 0
CARDIAC ENZYMES INCREASED (Investigations) | 4 | 1
CARDIAC STRESS TEST ABNORMAL (Investigations) | 1 | 2
COMPUTERISED TOMOGRAM ABNORMAL (Investigations) | 1 | 0
COMPUTERISED TOMOGRAM THORAX ABNORMAL (Investigations) | 1 | 0
EJECTION FRACTION DECREASED (Investigations) | 1 | 0
ELECTROCARDIOGRAM ST SEGMENT ELEVATION (Investigations) | 1 | 0
HAEMOGLOBIN DECREASED (Investigations) | 1 | 0
HEART RATE INCREASED (Investigations) | 1 | 0
OXYGEN CONSUMPTION INCREASED (Investigations) | 0 | 1
TROPONIN INCREASED (Investigations) | 2 | 0
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 7 | 5
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 5 | 1
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 6 | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 2
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 4 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 3 | 1
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 3 | 2
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 | 1
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 | 1
OBESITY (Metabolism and nutrition disorders) | 6 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 | 3
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 4 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 4
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 | 1
CHONDROCALCINOSIS PYROPHOSPHATE (Musculoskeletal and connective tissue disorders) | 1 | 0
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 2 | 0
DUPUYTREN'S CONTRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 1
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
FRACTURE NONUNION (Musculoskeletal and connective tissue disorders) | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 9 | 2
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1 | 0
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 7 | 2
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 4 | 0
MUSCULOSKELETAL DISORDER (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 3
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 26 | 14
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 | 2
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1 | 0
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 0
SACROILIITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 | 2
SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 3 | 2
TENDINOUS CONTRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0
VERTEBRAL FORAMINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ACUTE MYELOID LEUKAEMIA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
ADENOCARCINOMA PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-CELL LYMPHOMA STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
BENIGN OVARIAN TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BILE DUCT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
BLADDER CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
BLADDER CANCER STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
BREAST CANCER STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
GLIOBLASTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
HEAD AND NECK CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HEAD AND NECK CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HEPATIC CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HYPOPHARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LEUKAEMIA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LIP AND/OR ORAL CAVITY CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0
LUNG SQUAMOUS CELL CARCINOMA STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG SQUAMOUS CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO LYMPH NODES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO SPINE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ORAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OROPHARYNGEAL CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OVARIAN CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OVARIAN EPITHELIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
PERICARDIAL EFFUSION MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 3
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SINONASAL PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
SMALL CELL LUNG CANCER LIMITED STAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SMALL CELL LUNG CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
TONGUE NEOPLASM MALIGNANT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
URETERIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
VULVAL CANCER STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
APHASIA (Nervous system disorders) | 0 | 1
ARACHNOIDITIS (Nervous system disorders) | 0 | 1
AUTONOMIC NERVOUS SYSTEM IMBALANCE (Nervous system disorders) | 1 | 0
CAROTID ARTERY DISEASE (Nervous system disorders) | 2 | 0
CAROTID ARTERY STENOSIS (Nervous system disorders) | 11 | 7
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 1 | 0
CENTRAL NERVOUS SYSTEM LESION (Nervous system disorders) | 1 | 0
CEREBELLAR INFARCTION (Nervous system disorders) | 1 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 1 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 19 | 15
CEREBROVASCULAR DISORDER (Nervous system disorders) | 1 | 1
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 1 | 0
COMPLICATED MIGRAINE (Nervous system disorders) | 2 | 0
CONVULSION (Nervous system disorders) | 3 | 1
DIABETIC NEUROPATHY (Nervous system disorders) | 0 | 1
DIZZINESS (Nervous system disorders) | 6 | 1
DYSARTHRIA (Nervous system disorders) | 2 | 0
EMBOLIC STROKE (Nervous system disorders) | 1 | 0
ENCEPHALOPATHY (Nervous system disorders) | 2 | 2
GUILLAIN-BARRE SYNDROME (Nervous system disorders) | 2 | 0
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 | 1
HAEMORRHAGIC STROKE (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 2 | 3
HEMIPARESIS (Nervous system disorders) | 1 | 1
HEMIPLEGIC MIGRAINE (Nervous system disorders) | 1 | 0
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
HYPOAESTHESIA (Nervous system disorders) | 1 | 3
HYPOXIC-ISCHAEMIC ENCEPHALOPATHY (Nervous system disorders) | 2 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 5 | 3
LATERAL MEDULLARY SYNDROME (Nervous system disorders) | 1 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
LUMBAR RADICULOPATHY (Nervous system disorders) | 2 | 1
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 2 | 0
MIGRAINE (Nervous system disorders) | 2 | 1
MYELOMALACIA (Nervous system disorders) | 1 | 0
NEUROLOGICAL SYMPTOM (Nervous system disorders) | 1 | 0
NYSTAGMUS (Nervous system disorders) | 1 | 0
PARAESTHESIA (Nervous system disorders) | 4 | 1
POLYNEUROPATHY ALCOHOLIC (Nervous system disorders) | 1 | 0
POST-TRAUMATIC HEADACHE (Nervous system disorders) | 0 | 1
PRESYNCOPE (Nervous system disorders) | 5 | 1
RADICULITIS (Nervous system disorders) | 0 | 1
RADICULITIS CERVICAL (Nervous system disorders) | 1 | 0
SPONDYLITIC MYELOPATHY (Nervous system disorders) | 1 | 0
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 | 1
SUBDURAL HYGROMA (Nervous system disorders) | 2 | 0
SYNCOPE (Nervous system disorders) | 24 | 13
THALAMIC INFARCTION (Nervous system disorders) | 3 | 0
THROMBOTIC STROKE (Nervous system disorders) | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 11 | 6
UNRESPONSIVE TO STIMULI (Nervous system disorders) | 1 | 0
URAEMIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
VERTEBRAL ARTERY OCCLUSION (Nervous system disorders) | 0 | 1
VITH NERVE PARALYSIS (Nervous system disorders) | 2 | 1
ACUTE STRESS DISORDER (Psychiatric disorders) | 0 | 1
ADJUSTMENT DISORDER WITH MIXED DISTURBANCE OF EMOTION AND CONDUCT (Psychiatric disorders) | 0 | 1
ALCOHOL ABUSE (Psychiatric disorders) | 1 | 0
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 0 | 1
ANXIETY (Psychiatric disorders) | 2 | 1
BIPOLAR DISORDER (Psychiatric disorders) | 0 | 1
COMPLETED SUICIDE (Psychiatric disorders) | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 1
DELIRIUM (Psychiatric disorders) | 0 | 1
DELIRIUM TREMENS (Psychiatric disorders) | 0 | 1
DEPRESSION SUICIDAL (Psychiatric disorders) | 1 | 0
HALLUCINATION, VISUAL (Psychiatric disorders) | 0 | 1
INTENTIONAL SELF-INJURY (Psychiatric disorders) | 1 | 0
MAJOR DEPRESSION (Psychiatric disorders) | 2 | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 5 | 2
PANIC ATTACK (Psychiatric disorders) | 1 | 1
SUICIDAL IDEATION (Psychiatric disorders) | 0 | 2
CALCULUS URETERIC (Renal and urinary disorders) | 1 | 3
HAEMATURIA (Renal and urinary disorders) | 3 | 2
HYDRONEPHROSIS (Renal and urinary disorders) | 1 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 7 | 7
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 1 | 2
RENAL DISORDER (Renal and urinary disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 5 | 4
RENAL FAILURE ACUTE (Renal and urinary disorders) | 12 | 12
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 2 | 3
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 1
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 1 | 0
STRESS URINARY INCONTINENCE (Renal and urinary disorders) | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 4 | 1
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 3 | 3
FALLOPIAN TUBE CYST (Reproductive system and breast disorders) | 1 | 0
PELVIC HAEMATOMA (Reproductive system and breast disorders) | 1 | 0
UTERINE POLYP (Reproductive system and breast disorders) | 1 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 1
VULVA CYST (Reproductive system and breast disorders) | 1 | 0
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 4
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 16 | 7
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 2 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 28 | 10
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 33 | 13
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 5 | 3
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
HYPERVENTILATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 | 2
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
MEDIASTINAL MASS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
NASAL POLYPS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
NON-CARDIOGENIC PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ORGANISING PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 4 | 3
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 4
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 | 5
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 9 | 7
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 3 | 1
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 2 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 13 | 8
TRACHEAL STENOSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DIABETIC FOOT (Skin and subcutaneous tissue disorders) | 2 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 4 | 1
AORTIC ANEURYSM REPAIR (Surgical and medical procedures) | 1 | 0
CHOLECYSTECTOMY (Surgical and medical procedures) | 1 | 1
COLOSTOMY (Surgical and medical procedures) | 0 | 1
CORONARY ARTERY BYPASS (Surgical and medical procedures) | 1 | 0
HIP ARTHROPLASTY (Surgical and medical procedures) | 3 | 0
INGUINAL HERNIA REPAIR (Surgical and medical procedures) | 0 | 1
KNEE ARTHROPLASTY (Surgical and medical procedures) | 1 | 0
LEG AMPUTATION (Surgical and medical procedures) | 0 | 1
MEDICAL DEVICE REMOVAL (Surgical and medical procedures) | 0 | 1
NEPHRECTOMY (Surgical and medical procedures) | 1 | 0
SPINAL FUSION SURGERY (Surgical and medical procedures) | 1 | 0
TENDON OPERATION (Surgical and medical procedures) | 0 | 1
TRANSURETHRAL PROSTATECTOMY (Surgical and medical procedures) | 0 | 1
ACCELERATED HYPERTENSION (Vascular disorders) | 3 | 1
AORTIC ANEURYSM (Vascular disorders) | 6 | 2
AORTIC DISSECTION (Vascular disorders) | 0 | 1
AORTIC INTRAMURAL HAEMATOMA (Vascular disorders) | 1 | 1
AORTIC STENOSIS (Vascular disorders) | 4 | 5
ARTERIAL SPASM (Vascular disorders) | 1 | 0
ARTERIOSCLEROSIS (Vascular disorders) | 0 | 1
BLOOD PRESSURE INADEQUATELY CONTROLLED (Vascular disorders) | 1 | 0
CIRCULATORY COLLAPSE (Vascular disorders) | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 11 | 4
FEMORAL ARTERIAL STENOSIS (Vascular disorders) | 1 | 1
HAEMATOMA (Vascular disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 8 | 2
HYPERTENSIVE CRISIS (Vascular disorders) | 3 | 5
HYPOTENSION (Vascular disorders) | 5 | 4
ILIAC ARTERY STENOSIS (Vascular disorders) | 1 | 1
INTERMITTENT CLAUDICATION (Vascular disorders) | 8 | 7
MALIGNANT HYPERTENSION (Vascular disorders) | 1 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 2 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 3 | 8
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 | 1
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 7 | 6
SUBCLAVIAN ARTERY OCCLUSION (Vascular disorders) | 1 | 0
SUBCLAVIAN ARTERY STENOSIS (Vascular disorders) | 1 | 0
SUBCLAVIAN STEAL SYNDROME (Vascular disorders) | 1 | 0
THROMBOSIS (Vascular disorders) | 2 | 0
VASOSPAM (Vascular disorders) | 1 | 0
VENOUS INSUFFICIENCY (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Absorb BVS (N=1322) | XIENCE (N=686)
ANAEMIA (Blood and lymphatic system disorders) | 21 | 16
ANAEMIA OF CHRONIC DISEASE (Blood and lymphatic system disorders) | 1 | 1
COAGULOPATHY (Blood and lymphatic system disorders) | 0 | 2
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 2 | 4
HAEMORRHAGIC DIATHESIS (Blood and lymphatic system disorders) | 2 | 1
HEPARIN-INDUCED THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 3 | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 5 | 2
LYMPHADENITIS (Blood and lymphatic system disorders) | 1 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 2 | 0
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 2 | 0
NORMOCHROMIC NORMOCYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
SPLENIC INFARCTION (Blood and lymphatic system disorders) | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 2
ACUTE CORONARY SYNDROME (Cardiac disorders) | 6 | 5
ACUTE LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 49 | 22
ANGINA PECTORIS (Cardiac disorders) | 381 | 202
ANGINA UNSTABLE (Cardiac disorders) | 77 | 29
AORTIC VALVE DISEASE (Cardiac disorders) | 2 | 0
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 2 | 0
AORTIC VALVE STENOSIS (Cardiac disorders) | 8 | 2
ARRHYTHMIA (Cardiac disorders) | 1 | 3
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 4 | 0
ARTERIOSPASM CORONARY (Cardiac disorders) | 4 | 4
ATRIAL FIBRILLATION (Cardiac disorders) | 95 | 42
ATRIAL FLUTTER (Cardiac disorders) | 11 | 3
ATRIAL HYPERTROPHY (Cardiac disorders) | 0 | 1
ATRIAL TACHYCARDIA (Cardiac disorders) | 0 | 1
ATRIAL THROMBOSIS (Cardiac disorders) | 1 | 0
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 6 | 0
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 | 1
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 5 | 1
BRADYCARDIA (Cardiac disorders) | 31 | 13
BUNDLE BRANCH BLOCK (Cardiac disorders) | 0 | 1
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 0 | 1
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 1 | 1
CARDIAC ARREST (Cardiac disorders) | 10 | 6
CARDIAC FAILURE (Cardiac disorders) | 8 | 4
CARDIAC FAILURE ACUTE (Cardiac disorders) | 5 | 1
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 2 | 3
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 39 | 30
CARDIAC FLUTTER (Cardiac disorders) | 2 | 1
CARDIAC TAMPONADE (Cardiac disorders) | 1 | 0
CARDIAC VALVE DISEASE (Cardiac disorders) | 2 | 0
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 2 | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 1 | 3
CARDIOMEGALY (Cardiac disorders) | 1 | 0
CARDIOMYOPATHY (Cardiac disorders) | 1 | 2
CARDIORENAL SYNDROME (Cardiac disorders) | 1 | 0
CHRONIC LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1 | 0
CONDUCTION DISORDER (Cardiac disorders) | 0 | 1
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 44 | 28
CORONARY ARTERY DISSECTION (Cardiac disorders) | 85 | 56
CORONARY ARTERY EMBOLISM (Cardiac disorders) | 3 | 4
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 5 | 2
CORONARY ARTERY PERFORATION (Cardiac disorders) | 7 | 3
CORONARY ARTERY STENOSIS (Cardiac disorders) | 23 | 14
CORONARY NO-REFLOW PHENOMENON (Cardiac disorders) | 1 | 1
CORONARY OSTIAL STENOSIS (Cardiac disorders) | 1 | 0
CYANOSIS (Cardiac disorders) | 0 | 1
DIASTOLIC DYSFUNCTION (Cardiac disorders) | 1 | 0
DRESSLER'S SYNDROME (Cardiac disorders) | 0 | 3
EXTRASYSTOLES (Cardiac disorders) | 1 | 1
HEART VALVE INCOMPETENCE (Cardiac disorders) | 1 | 0
HYPERTROPHIC CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
IN-STENT CORONARY ARTERY RESTENOSIS (Cardiac disorders) | 4 | 5
INTRACARDIAC THROMBUS (Cardiac disorders) | 1 | 1
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 4 | 2
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 | 1
LEFT VENTRICULAR HYPERTROPHY (Cardiac disorders) | 1 | 0
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 8 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 54 | 24
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 6 | 1
NODAL ARRHYTHMIA (Cardiac disorders) | 0 | 1
NODAL RHYTHM (Cardiac disorders) | 1 | 0
PALPITATIONS (Cardiac disorders) | 32 | 17
PERICARDIAL EFFUSION (Cardiac disorders) | 6 | 3
PERICARDITIS (Cardiac disorders) | 1 | 1
PRINZMETAL ANGINA (Cardiac disorders) | 2 | 0
SICK SINUS SYNDROME (Cardiac disorders) | 6 | 4
SINUS ARREST (Cardiac disorders) | 1 | 0
SINUS ARRHYTHMIA (Cardiac disorders) | 0 | 1
SINUS BRADYCARDIA (Cardiac disorders) | 3 | 3
SINUS TACHYCARDIA (Cardiac disorders) | 2 | 0
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 12 | 5
TACHYCARDIA (Cardiac disorders) | 12 | 6
TORSADE DE POINTES (Cardiac disorders) | 1 | 0
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 2 | 0
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 | 1
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 6 | 0
VENTRICULAR FIBRILLATION (Cardiac disorders) | 6 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 14 | 6
ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 1 | 1
CYSTIC LYMPHANGIOMA (Congenital, familial and genetic disorders) | 1 | 0
MYOTONIC DYSTROPHY (Congenital, familial and genetic disorders) | 1 | 0
PULMONARY ARTERIOVENOUS FISTULA (Congenital, familial and genetic disorders) | 0 | 1
DEAFNESS (Ear and labyrinth disorders) | 1 | 1
EAR PAIN (Ear and labyrinth disorders) | 0 | 2
EUSTACHIAN TUBE OBSTRUCTION (Ear and labyrinth disorders) | 1 | 0
MIXED DEAFNESS (Ear and labyrinth disorders) | 1 | 0
TINNITUS (Ear and labyrinth disorders) | 1 | 2
TYMPANIC MEMBRANE PERFORATION (Ear and labyrinth disorders) | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 13 | 7
ADRENAL MASS (Endocrine disorders) | 1 | 0
GOITRE (Endocrine disorders) | 1 | 0
HYPERTHYROIDISM (Endocrine disorders) | 0 | 1
HYPOGONADISM (Endocrine disorders) | 0 | 1
HYPOTHYROIDISM (Endocrine disorders) | 6 | 1
THYROID CYST (Endocrine disorders) | 1 | 0
AGE-RELATED MACULAR DEGENERATION (Eye disorders) | 1 | 0
AMAUROSIS FUGAX (Eye disorders) | 1 | 0
CATARACT (Eye disorders) | 7 | 8
CATARACT NUCLEAR (Eye disorders) | 1 | 0
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 2 | 0
CONJUNCTIVITIS (Eye disorders) | 2 | 2
DIABETIC RETINOPATHY (Eye disorders) | 1 | 0
DIPLOPIA (Eye disorders) | 1 | 0
EYE PRURITUS (Eye disorders) | 1 | 0
EYE SWELLING (Eye disorders) | 0 | 1
GAZE PALSY (Eye disorders) | 1 | 0
GLAUCOMA (Eye disorders) | 4 | 0
MACULAR FIBROSIS (Eye disorders) | 1 | 0
MACULAR OEDEMA (Eye disorders) | 1 | 0
PAPILLOEDEMA (Eye disorders) | 1 | 0
POSTERIOR CAPSULE OPACIFICATION (Eye disorders) | 1 | 0
RETINAL DETACHMENT (Eye disorders) | 2 | 1
RETINAL HAEMORRHAGE (Eye disorders) | 1 | 1
SCLERAL DISCOLOURATION (Eye disorders) | 1 | 0
SCLERAL HAEMORRHAGE (Eye disorders) | 1 | 0
VISION BLURRED (Eye disorders) | 5 | 1
VISUAL IMPAIRMENT (Eye disorders) | 2 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 5 | 4
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 1
ABDOMINAL HERNIA (Gastrointestinal disorders) | 3 | 3
ABDOMINAL HERNIA OBSTRUCTIVE (Gastrointestinal disorders) | 1 | 0
ABDOMINAL MASS (Gastrointestinal disorders) | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 13 | 13
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 8 | 7
ABDOMINAL WALL HAEMATOMA (Gastrointestinal disorders) | 1 | 0
ALCOHOLIC PANCREATITIS (Gastrointestinal disorders) | 0 | 1
BARRETT'S OESOPHAGUS (Gastrointestinal disorders) | 3 | 0
COELIAC ARTERY STENOSIS (Gastrointestinal disorders) | 1 | 0
COELIAC DISEASE (Gastrointestinal disorders) | 0 | 1
COLITIS (Gastrointestinal disorders) | 4 | 3
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 1 | 1
COLONIC POLYP (Gastrointestinal disorders) | 3 | 1
CONSTIPATION (Gastrointestinal disorders) | 11 | 2
CROHN'S DISEASE (Gastrointestinal disorders) | 2 | 1
DENTAL CARIES (Gastrointestinal disorders) | 1 | 0
DIABETIC GASTROPARESIS (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 18 | 7
DIVERTICULUM (Gastrointestinal disorders) | 3 | 1
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 1 | 1
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 2 | 1
DRY MOUTH (Gastrointestinal disorders) | 1 | 0
DUODENAL ULCER (Gastrointestinal disorders) | 1 | 0
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
DUODENITIS (Gastrointestinal disorders) | 2 | 0
DYSPEPSIA (Gastrointestinal disorders) | 15 | 4
DYSPHAGIA (Gastrointestinal disorders) | 10 | 2
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 1 | 0
EROSIVE OESOPHAGITIS (Gastrointestinal disorders) | 1 | 0
ERUCTATION (Gastrointestinal disorders) | 0 | 1
FAECAL INCONTINENCE (Gastrointestinal disorders) | 1 | 0
FAECALOMA (Gastrointestinal disorders) | 1 | 0
FAECES DISCOLOURED (Gastrointestinal disorders) | 1 | 1
FLATULENCE (Gastrointestinal disorders) | 2 | 0
FOOD POISONING (Gastrointestinal disorders) | 1 | 0
FUNCTIONAL GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1 | 0
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 2 | 4
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 2 | 0
GASTRITIS (Gastrointestinal disorders) | 6 | 3
GASTRITIS EROSIVE (Gastrointestinal disorders) | 3 | 0
GASTROINTESTINAL ANGIODYSPLASIA (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 2 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 16 | 15
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 23 | 8
HAEMATEMESIS (Gastrointestinal disorders) | 2 | 2
HAEMATOCHEZIA (Gastrointestinal disorders) | 4 | 0
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 4 | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0
HIATUS HERNIA (Gastrointestinal disorders) | 9 | 4
HYPOAESTHESIA ORAL (Gastrointestinal disorders) | 1 | 0
ILEUS (Gastrointestinal disorders) | 1 | 2
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 3 | 1
INFREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 1 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 4 | 6
INTESTINAL MASS (Gastrointestinal disorders) | 2 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 2
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 2 | 0
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 3 | 2
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 1 | 0
MELAENA (Gastrointestinal disorders) | 2 | 1
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 2 | 0
MOUTH ULCERATION (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 19 | 13
OESOPHAGEAL ACHALASIA (Gastrointestinal disorders) | 0 | 1
OESOPHAGEAL FOOD IMPACTION (Gastrointestinal disorders) | 1 | 0
OESOPHAGEAL PAIN (Gastrointestinal disorders) | 1 | 0
OESOPHAGEAL SPASM (Gastrointestinal disorders) | 1 | 1
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 1 | 0
OESOPHAGITIS (Gastrointestinal disorders) | 2 | 0
PANCREATIC CYST (Gastrointestinal disorders) | 1 | 3
PANCREATITIS (Gastrointestinal disorders) | 1 | 3
PANCREATITIS ACUTE (Gastrointestinal disorders) | 2 | 1
PANCREATITIS CHRONIC (Gastrointestinal disorders) | 1 | 0
PEPTIC ULCER (Gastrointestinal disorders) | 1 | 0
PROCTALGIA (Gastrointestinal disorders) | 1 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 8 | 8
RECTAL PROLAPSE (Gastrointestinal disorders) | 0 | 1
RETROPERITONEAL HAEMATOMA (Gastrointestinal disorders) | 2 | 0
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 | 6
SMALL INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 1 | 0
TONGUE CYST (Gastrointestinal disorders) | 1 | 0
TONGUE HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
TOOTH SOCKET HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
UMBILICAL HERNIA (Gastrointestinal disorders) | 4 | 2
UMBILICAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 2 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 3 | 4
VOMITING (Gastrointestinal disorders) | 13 | 10
ABASIA (General disorders) | 0 | 1
ADVERSE DRUG REACTION (General disorders) | 74 | 42
ASTHENIA (General disorders) | 12 | 4
BREAST COMPLICATION ASSOCIATED WITH DEVICE (General disorders) | 0 | 1
CARDIAC DEATH (General disorders) | 1 | 0
CATHETER SITE HAEMATOMA (General disorders) | 30 | 14
CATHETER SITE HAEMORRHAGE (General disorders) | 22 | 14
CATHETER SITE PAIN (General disorders) | 29 | 15
CATHETER SITE RASH (General disorders) | 0 | 1
CATHETER SITE RELATED REACTION (General disorders) | 9 | 4
CATHETER SITE SWELLING (General disorders) | 5 | 2
CHEST DISCOMFORT (General disorders) | 87 | 34
CHEST PAIN (General disorders) | 79 | 49
CHILLS (General disorders) | 0 | 1
CYST (General disorders) | 1 | 1
DEATH (General disorders) | 10 | 6
DEVICE ELECTRICAL FINDING (General disorders) | 0 | 1
DEVICE FAILURE (General disorders) | 1 | 1
DEVICE MALFUNCTION (General disorders) | 1 | 0
DEVICE OCCLUSION (General disorders) | 1 | 0
DISCOMFORT (General disorders) | 1 | 1
DROWNING (General disorders) | 1 | 0
DRUG INTOLERANCE (General disorders) | 2 | 0
DRUG WITHDRAWAL SYNDROME (General disorders) | 1 | 0
FACE OEDEMA (General disorders) | 0 | 1
FATIGUE (General disorders) | 50 | 20
FEELING COLD (General disorders) | 0 | 1
GAIT DISTURBANCE (General disorders) | 1 | 1
GENERALISED OEDEMA (General disorders) | 1 | 0
HERNIA (General disorders) | 0 | 1
HERNIA OBSTRUCTIVE (General disorders) | 1 | 0
HERNIA PAIN (General disorders) | 0 | 1
IMPAIRED HEALING (General disorders) | 0 | 2
IMPLANT SITE HAEMORRHAGE (General disorders) | 1 | 0
IMPLANT SITE PAIN (General disorders) | 1 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 2 | 1
LOCAL SWELLING (General disorders) | 2 | 0
MALAISE (General disorders) | 3 | 1
MASS (General disorders) | 1 | 1
MEDICAL DEVICE SITE REACTION (General disorders) | 1 | 0
MULTI-ORGAN FAILURE (General disorders) | 1 | 2
NON-CARDIAC CHEST PAIN (General disorders) | 271 | 122
OEDEMA (General disorders) | 2 | 0
OEDEMA PERIPHERAL (General disorders) | 25 | 10
PAIN (General disorders) | 9 | 6
PELVIC MASS (General disorders) | 0 | 2
PYREXIA (General disorders) | 9 | 3
SPINAL PAIN (General disorders) | 1 | 0
SUDDEN CARDIAC DEATH (General disorders) | 0 | 1
SURGICAL FAILURE (General disorders) | 1 | 0
SWELLING (General disorders) | 1 | 0
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 3 | 1
THROMBOSIS IN DEVICE (General disorders) | 14 | 6
BILE DUCT STONE (Hepatobiliary disorders) | 2 | 0
BILIARY COLIC (Hepatobiliary disorders) | 0 | 1
CHOLANGITIS (Hepatobiliary disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 4 | 2
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 2 | 4
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 12 | 6
GALLBLADDER DISORDER (Hepatobiliary disorders) | 1 | 0
HEPATIC LESION (Hepatobiliary disorders) | 2 | 1
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 | 0
HEPATOMEGALY (Hepatobiliary disorders) | 0 | 1
ISCHAEMIC HEPATITIS (Hepatobiliary disorders) | 1 | 0
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 1 | 0
ALLERGY TO ARTHROPOD STING (Immune system disorders) | 1 | 1
ANAPHYLACTIC REACTION (Immune system disorders) | 1 | 0
CONTRAST MEDIA ALLERGY (Immune system disorders) | 2 | 2
DRUG HYPERSENSITIVITY (Immune system disorders) | 5 | 4
FOOD ALLERGY (Immune system disorders) | 2 | 0
HYPERSENSITIVITY (Immune system disorders) | 0 | 2
SEASONAL ALLERGY (Immune system disorders) | 1 | 1
ABDOMINAL ABSCESS (Infections and infestations) | 0 | 1
ABDOMINAL INFECTION (Infections and infestations) | 1 | 0
ABSCESS NECK (Infections and infestations) | 1 | 0
ACUTE SINUSITIS (Infections and infestations) | 3 | 1
ACUTE TONSILLITIS (Infections and infestations) | 1 | 0
APPENDICITIS (Infections and infestations) | 4 | 2
APPENDICITIS PERFORATED (Infections and infestations) | 1 | 0
ARTERIOVENOUS GRAFT SITE INFECTION (Infections and infestations) | 0 | 1
ARTHRITIS BACTERIAL (Infections and infestations) | 1 | 0
ARTHRITIS INFECTIVE (Infections and infestations) | 1 | 0
BACTERAEMIA (Infections and infestations) | 4 | 0
BACTERIAL DISEASE CARRIER (Infections and infestations) | 0 | 1
BACTERIAL INFECTION (Infections and infestations) | 0 | 1
BACTERIAL SEPSIS (Infections and infestations) | 0 | 2
BREAST ABSCESS (Infections and infestations) | 0 | 1
BREAST CELLULITIS (Infections and infestations) | 1 | 0
BRONCHITIS (Infections and infestations) | 34 | 21
BRONCHITIS VIRAL (Infections and infestations) | 1 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 1
CARBUNCLE (Infections and infestations) | 0 | 1
CATHETER SITE ABSCESS (Infections and infestations) | 2 | 0
CATHETER SITE CELLULITIS (Infections and infestations) | 3 | 0
CATHETER SITE INFECTION (Infections and infestations) | 1 | 1
CELLULITIS (Infections and infestations) | 15 | 14
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 0 | 2
CLOSTRIDIAL INFECTION (Infections and infestations) | 4 | 1
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 3 | 3
CYSTITIS (Infections and infestations) | 2 | 1
DIABETIC FOOT INFECTION (Infections and infestations) | 1 | 0
DIVERTICULITIS (Infections and infestations) | 5 | 3
EAR INFECTION (Infections and infestations) | 3 | 0
ENDOCARDITIS (Infections and infestations) | 1 | 0
ENTEROCOCCAL SEPSIS (Infections and infestations) | 0 | 1
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 | 0
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
EYELID INFECTION (Infections and infestations) | 1 | 0
FOLLICULITIS (Infections and infestations) | 1 | 0
FUNGAL INFECTION (Infections and infestations) | 0 | 1
FURUNCLE (Infections and infestations) | 1 | 0
GANGRENE (Infections and infestations) | 1 | 1
GASTROENTERITIS (Infections and infestations) | 10 | 3
GASTROENTERITIS VIRAL (Infections and infestations) | 4 | 3
GENITAL INFECTION FEMALE (Infections and infestations) | 1 | 0
GROIN ABSCESS (Infections and infestations) | 1 | 0
HELICOBACTER INFECTION (Infections and infestations) | 2 | 0
HEPATITIS C (Infections and infestations) | 2 | 0
HERPES ZOSTER (Infections and infestations) | 7 | 3
HERPES ZOSTER OPHTHALMIC (Infections and infestations) | 1 | 0
HIV INFECTION (Infections and infestations) | 1 | 0
IMPLANT SITE INFECTION (Infections and infestations) | 1 | 0
INFECTED DERMAL CYST (Infections and infestations) | 1 | 0
INFECTED SKIN ULCER (Infections and infestations) | 0 | 1
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 1 | 0
INFLUENZA (Infections and infestations) | 8 | 8
KIDNEY INFECTION (Infections and infestations) | 4 | 0
LARYNGITIS (Infections and infestations) | 2 | 1
LOBAR PNEUMONIA (Infections and infestations) | 3 | 1
LOCALISED INFECTION (Infections and infestations) | 0 | 3
LUNG ABSCESS (Infections and infestations) | 0 | 1
MENINGITIS ASEPTIC (Infections and infestations) | 1 | 0
METAPNEUMOVIRUS INFECTION (Infections and infestations) | 1 | 0
MYCOBACTERIUM ABSCESSUS INFECTION (Infections and infestations) | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 6 | 5
ONYCHOMYCOSIS (Infections and infestations) | 2 | 0
ORAL FUNGAL INFECTION (Infections and infestations) | 1 | 0
ORCHITIS (Infections and infestations) | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 3 | 4
OTITIS EXTERNA (Infections and infestations) | 1 | 1
OTITIS MEDIA (Infections and infestations) | 1 | 0
OTITIS MEDIA ACUTE (Infections and infestations) | 1 | 0
PARONYCHIA (Infections and infestations) | 2 | 0
PERITONITIS (Infections and infestations) | 0 | 1
PERITONSILLAR ABSCESS (Infections and infestations) | 1 | 0
PHARYNGITIS (Infections and infestations) | 1 | 0
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 | 1
PILONIDAL CYST (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 33 | 27
PNEUMONIA ADENOVIRAL (Infections and infestations) | 1 | 0
PNEUMONIA BACTERIAL (Infections and infestations) | 2 | 0
PNEUMONIA NECROTISING (Infections and infestations) | 1 | 0
PNEUMONIA PRIMARY ATYPICAL (Infections and infestations) | 1 | 0
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 2 | 0
POST PROCEDURAL CELLULITIS (Infections and infestations) | 1 | 0
POST PROCEDURAL INFECTION (Infections and infestations) | 3 | 0
POST PROCEDURAL PNEUMONIA (Infections and infestations) | 1 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 | 1
PROSTATE INFECTION (Infections and infestations) | 1 | 0
PYELONEPHRITIS (Infections and infestations) | 1 | 0
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1
SEPSIS (Infections and infestations) | 15 | 10
SEPSIS SYNDROME (Infections and infestations) | 2 | 0
SEPTIC ENCEPHALOPATHY (Infections and infestations) | 0 | 1
SEPTIC SHOCK (Infections and infestations) | 2 | 1
SINUSITIS (Infections and infestations) | 11 | 10
SPINAL CORD INFECTION (Infections and infestations) | 1 | 0
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 2
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 | 0
TINEA PEDIS (Infections and infestations) | 1 | 0
TOOTH ABSCESS (Infections and infestations) | 2 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 25 | 6
URINARY TRACT INFECTION (Infections and infestations) | 32 | 23
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 1 | 1
UROSEPSIS (Infections and infestations) | 3 | 4
VIRAL INFECTION (Infections and infestations) | 4 | 3
VIRAL LABYRINTHITIS (Infections and infestations) | 0 | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 2
WOUND INFECTION (Infections and infestations) | 2 | 3
WOUND INFECTION BACTERIAL (Infections and infestations) | 0 | 1
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1 | 2
ACCIDENT (Injury, poisoning and procedural complications) | 0 | 1
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 2 | 0
ACETABULUM FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 3 | 2
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 5 | 3
ANIMAL BITE (Injury, poisoning and procedural complications) | 2 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 4
ANXIETY POSTOPERATIVE (Injury, poisoning and procedural complications) | 1 | 1
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 2 | 0
ARTHROPOD STING (Injury, poisoning and procedural complications) | 1 | 1
ASBESTOSIS (Injury, poisoning and procedural complications) | 1 | 0
AVULSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
BURNS THIRD DEGREE (Injury, poisoning and procedural complications) | 1 | 1
CARDIAC FUNCTION DISTURBANCE POSTOPERATIVE (Injury, poisoning and procedural complications) | 0 | 1
CARDIAC PROCEDURE COMPLICATION (Injury, poisoning and procedural complications) | 4 | 4
CATHETER SITE HAEMATOMA (Injury, poisoning and procedural complications) | 10 | 8
CEREBRAL HAEMORRHAGE TRAUMATIC (Injury, poisoning and procedural complications) | 2 | 0
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
COLON INJURY (Injury, poisoning and procedural complications) | 1 | 0
CONCUSSION (Injury, poisoning and procedural complications) | 1 | 1
CONTRAST MEDIA ALLERGY (Injury, poisoning and procedural complications) | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 25 | 6
CORNEAL ABRASION (Injury, poisoning and procedural complications) | 0 | 1
CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 51 | 15
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 3 | 1
CYSTITIS RADIATION (Injury, poisoning and procedural complications) | 1 | 0
DEEP VEIN THROMBOSIS POSTOPERATIVE (Injury, poisoning and procedural complications) | 2 | 0
DRUG ADMINISTRATION ERROR (Injury, poisoning and procedural complications) | 1 | 0
EXCORIATION (Injury, poisoning and procedural complications) | 2 | 0
EXPOSURE TO TOXIC AGENT (Injury, poisoning and procedural complications) | 2 | 0
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
FALL (Injury, poisoning and procedural complications) | 28 | 20
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 | 2
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 3 | 0
FOOT FRACTURE (Injury, poisoning and procedural complications) | 4 | 1
FOREIGN BODY (Injury, poisoning and procedural complications) | 0 | 1
GASTROINTESTINAL ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 0 | 1
HAEMATURIA TRAUMATIC (Injury, poisoning and procedural complications) | 1 | 0
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
HEAD INJURY (Injury, poisoning and procedural complications) | 1 | 2
HIP FRACTURE (Injury, poisoning and procedural complications) | 4 | 2
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 3 | 2
ILIOTIBIAL BAND SYNDROME (Injury, poisoning and procedural complications) | 0 | 1
IN-STENT ARTERIAL RESTENOSIS (Injury, poisoning and procedural complications) | 0 | 1
IN-STENT CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 8 | 6
INCISION SITE PRURITUS (Injury, poisoning and procedural complications) | 0 | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 3 | 0
INJURY (Injury, poisoning and procedural complications) | 2 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 | 1
JOINT INJURY (Injury, poisoning and procedural complications) | 2 | 0
LACERATION (Injury, poisoning and procedural complications) | 7 | 4
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 | 6
LIMB INJURY (Injury, poisoning and procedural complications) | 3 | 4
LIMB TRAUMATIC AMPUTATION (Injury, poisoning and procedural complications) | 1 | 0
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
MENISCUS LESION (Injury, poisoning and procedural complications) | 8 | 4
MOUTH INJURY (Injury, poisoning and procedural complications) | 0 | 1
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 2 | 0
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 1 | 0
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 0 | 1
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 2 | 1
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
PERIORBITAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
PLAQUE SHIFT (Injury, poisoning and procedural complications) | 4 | 6
POST CONCUSSION SYNDROME (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL CONSTIPATION (Injury, poisoning and procedural complications) | 0 | 1
POST PROCEDURAL DISCOMFORT (Injury, poisoning and procedural complications) | 0 | 1
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 3 | 2
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 6 | 4
POST PROCEDURAL MYOCARDIAL INFARCTION (Injury, poisoning and procedural complications) | 12 | 7
POST PROCEDURAL STROKE (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL SWELLING (Injury, poisoning and procedural complications) | 0 | 1
POST-TRAUMATIC NECK SYNDROME (Injury, poisoning and procedural complications) | 0 | 1
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 4 | 1
POSTOPERATIVE ADHESION (Injury, poisoning and procedural complications) | 1 | 0
POSTOPERATIVE FEVER (Injury, poisoning and procedural complications) | 1 | 0
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 2 | 0
PROCEDURAL DIZZINESS (Injury, poisoning and procedural complications) | 1 | 2
PROCEDURAL HEADACHE (Injury, poisoning and procedural complications) | 5 | 2
PROCEDURAL HYPERTENSION (Injury, poisoning and procedural complications) | 10 | 4
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 13 | 7
PROCEDURAL NAUSEA (Injury, poisoning and procedural complications) | 8 | 4
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 3 | 3
PROCEDURAL VOMITING (Injury, poisoning and procedural complications) | 3 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
RESPIRATORY FUME INHALATION DISORDER (Injury, poisoning and procedural complications) | 1 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 4 | 3
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 10 | 2
SCAPULA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
SEROMA (Injury, poisoning and procedural complications) | 1 | 0
SKULL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
SNAKE BITE (Injury, poisoning and procedural complications) | 1 | 0
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 1 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 6 | 2
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 2 | 1
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 6 | 4
SUTURE RELATED COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1
TENDON INJURY (Injury, poisoning and procedural complications) | 0 | 2
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 | 2
THERMAL BURN (Injury, poisoning and procedural complications) | 1 | 0
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 | 4
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 | 1
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 5 | 2
TRAUMATIC HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1
ULNA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 4 | 0
URINARY RETENTION POSTOPERATIVE (Injury, poisoning and procedural complications) | 5 | 1
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
VASCULAR GRAFT OCCLUSION (Injury, poisoning and procedural complications) | 2 | 1
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 10 | 6
WOUND (Injury, poisoning and procedural complications) | 1 | 0
WOUND EVISCERATION (Injury, poisoning and procedural complications) | 1 | 0
WOUND HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 1
WRIST FRACTURE (Injury, poisoning and procedural complications) | 3 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
ANGIOGRAM (Investigations) | 1 | 0
ARTERIOGRAM CORONARY ABNORMAL (Investigations) | 1 | 2
BIOPSY LUNG (Investigations) | 0 | 1
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 3 | 0
BLOOD CREATINE INCREASED (Investigations) | 1 | 0
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 12 | 8
BLOOD CREATINE PHOSPHOKINASE MB INCREASED (Investigations) | 153 | 72
BLOOD CREATININE INCREASED (Investigations) | 5 | 2
BLOOD GLUCOSE DECREASED (Investigations) | 0 | 1
BLOOD GLUCOSE INCREASED (Investigations) | 4 | 1
BLOOD HOMOCYSTEINE INCREASED (Investigations) | 1 | 0
BLOOD IRON DECREASED (Investigations) | 0 | 1
BLOOD MAGNESIUM DECREASED (Investigations) | 0 | 1
BLOOD POTASSIUM DECREASED (Investigations) | 1 | 0
BLOOD PRESSURE DECREASED (Investigations) | 0 | 1
BLOOD PRESSURE INCREASED (Investigations) | 12 | 4
BLOOD PRESSURE ORTHOSTATIC ABNORMAL (Investigations) | 1 | 0
BLOOD PRESSURE SYSTOLIC INCREASED (Investigations) | 1 | 0
BLOOD TESTOSTERONE DECREASED (Investigations) | 0 | 1
BLOOD THYROID STIMULATING HORMONE DECREASED (Investigations) | 1 | 0
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 3 | 0
BLOOD URIC ACID INCREASED (Investigations) | 0 | 1
BLOOD URINE PRESENT (Investigations) | 1 | 0
BONE DENSITY ABNORMAL (Investigations) | 0 | 1
BREATH SOUNDS ABNORMAL (Investigations) | 0 | 1
CARDIAC ENZYMES INCREASED (Investigations) | 104 | 45
CARDIAC MURMUR (Investigations) | 1 | 0
CARDIAC STRESS TEST ABNORMAL (Investigations) | 9 | 3
CAROTID BRUIT (Investigations) | 7 | 3
CATHETERISATION CARDIAC (Investigations) | 0 | 1
CLOSTRIDIUM TEST POSITIVE (Investigations) | 1 | 0
COMPUTERISED TOMOGRAM ABNORMAL (Investigations) | 1 | 0
COMPUTERISED TOMOGRAM THORAX ABNORMAL (Investigations) | 1 | 0
ECHOCARDIOGRAM ABNORMAL (Investigations) | 1 | 0
EJECTION FRACTION ABNORMAL (Investigations) | 1 | 0
EJECTION FRACTION DECREASED (Investigations) | 1 | 0
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 0 | 1
ELECTROCARDIOGRAM CHANGE (Investigations) | 4 | 1
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 | 1
ELECTROCARDIOGRAM ST SEGMENT ABNORMAL (Investigations) | 0 | 1
ELECTROCARDIOGRAM ST SEGMENT ELEVATION (Investigations) | 8 | 0
ELECTROCARDIOGRAM ST-T CHANGE (Investigations) | 1 | 0
FEMORAL BRUIT (Investigations) | 0 | 1
GLOMERULAR FILTRATION RATE DECREASED (Investigations) | 1 | 0
GLYCOSYLATED HAEMOGLOBIN INCREASED (Investigations) | 1 | 1
HAEMOGLOBIN DECREASED (Investigations) | 3 | 0
HEART RATE DECREASED (Investigations) | 1 | 0
HEART RATE INCREASED (Investigations) | 4 | 0
HEART RATE IRREGULAR (Investigations) | 1 | 2
HELICOBACTER TEST POSITIVE (Investigations) | 0 | 1
HEPATIC ENZYME INCREASED (Investigations) | 4 | 1
LIPIDS ABNORMAL (Investigations) | 0 | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 2 | 4
METABOLIC FUNCTION TEST ABNORMAL (Investigations) | 1 | 0
OCCULT BLOOD POSITIVE (Investigations) | 2 | 0
OXYGEN CONSUMPTION INCREASED (Investigations) | 0 | 1
PROSTATIC SPECIFIC ANTIGEN INCREASED (Investigations) | 2 | 0
RED BLOOD CELL COUNT DECREASED (Investigations) | 0 | 1
RED BLOOD CELL SEDIMENTATION RATE INCREASED (Investigations) | 0 | 1
RENAL FUNCTION TEST ABNORMAL (Investigations) | 2 | 0
THYROID FUNCTION TEST ABNORMAL (Investigations) | 1 | 0
TROPONIN I INCREASED (Investigations) | 24 | 10
TROPONIN INCREASED (Investigations) | 50 | 20
TROPONIN T INCREASED (Investigations) | 0 | 1
URINE LEUKOCYTE ESTERASE POSITIVE (Investigations) | 1 | 0
VITAMIN B12 DECREASED (Investigations) | 1 | 0
VITAMIN D DECREASED (Investigations) | 1 | 1
WEIGHT DECREASED (Investigations) | 3 | 1
WEIGHT INCREASED (Investigations) | 4 | 0
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 2 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 11 | 11
DIABETES MELLITUS (Metabolism and nutrition disorders) | 9 | 3
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1 | 0
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 5 | 1
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 2 | 2
FLUID RETENTION (Metabolism and nutrition disorders) | 1 | 0
GOUT (Metabolism and nutrition disorders) | 5 | 2
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 14 | 7
HYPERKALAEMIA (Metabolism and nutrition disorders) | 4 | 5
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPERURICAEMIA (Metabolism and nutrition disorders) | 2 | 0
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 10 | 3
HYPOKALAEMIA (Metabolism and nutrition disorders) | 15 | 11
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 5 | 3
HYPONATRAEMIA (Metabolism and nutrition disorders) | 8 | 5
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1 | 1
IMPAIRED FASTING GLUCOSE (Metabolism and nutrition disorders) | 1 | 0
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 | 1
OBESITY (Metabolism and nutrition disorders) | 6 | 3
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 5 | 4
VITAMIN B COMPLEX DEFICIENCY (Metabolism and nutrition disorders) | 1 | 0
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 27 | 16
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 8 | 5
ARTHROFIBROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 55 | 28
BONE LESION (Musculoskeletal and connective tissue disorders) | 0 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
BURSITIS (Musculoskeletal and connective tissue disorders) | 4 | 4
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
CHONDROCALCINOSIS PYROPHOSPHATE (Musculoskeletal and connective tissue disorders) | 1 | 0
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 6 | 1
DUPUYTREN'S CONTRACTURE (Musculoskeletal and connective tissue disorders) | 2 | 1
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 0 | 2
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 3
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 | 1
FRACTURE NONUNION (Musculoskeletal and connective tissue disorders) | 1 | 0
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 2 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 9 | 2
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1 | 0
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 4 | 1
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 3 | 2
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 7 | 2
MOBILITY DECREASED (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 10 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 6 | 4
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 21 | 7
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 5 | 2
MUSCULOSKELETAL DISORDER (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 18 | 16
MYALGIA (Musculoskeletal and connective tissue disorders) | 12 | 8
MYOSITIS (Musculoskeletal and connective tissue disorders) | 2 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 7 | 5
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 30 | 18
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 40 | 15
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 7 | 1
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
PLANTAR FASCIITIS (Musculoskeletal and connective tissue disorders) | 2 | 1
POLYMYALGIA RHEUMATICA (Musculoskeletal and connective tissue disorders) | 0 | 2
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 0
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 8 | 4
SACROILIITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 6 | 4
SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 3 | 2
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 1 | 1
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 0 | 1
TENDINOUS CONTRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
TENOSYNOVITIS STENOSANS (Musculoskeletal and connective tissue disorders) | 0 | 1
TRIGGER FINGER (Musculoskeletal and connective tissue disorders) | 1 | 0
VERTEBRAL FORAMINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
ACOUSTIC NEUROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ACUTE MYELOID LEUKAEMIA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
ADENOCARCINOMA PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-CELL LYMPHOMA STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 7
BENIGN BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BENIGN OVARIAN TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BILE DUCT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
BLADDER CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
BLADDER CANCER STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
BREAST CANCER STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
GLIOBLASTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
HAEMANGIOMA OF SPLEEN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
HEAD AND NECK CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HEAD AND NECK CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HEPATIC CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HYPOPHARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LEUKAEMIA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LIP AND/OR ORAL CAVITY CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 6
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 0
LUNG SQUAMOUS CELL CARCINOMA STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG SQUAMOUS CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO LYMPH NODES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO SPINE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
NEURILEMMOMA MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ORAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OROPHARYNGEAL CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OVARIAN CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OVARIAN EPITHELIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
PERICARDIAL EFFUSION MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 4
PROSTATE CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RENAL HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
SINONASAL PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SMALL CELL LUNG CANCER LIMITED STAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SMALL CELL LUNG CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
TONGUE NEOPLASM MALIGNANT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
URETERIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
VULVAL CANCER STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
AMNESIA (Nervous system disorders) | 4 | 2
APHASIA (Nervous system disorders) | 0 | 1
ARACHNOIDITIS (Nervous system disorders) | 0 | 1
ATAXIA (Nervous system disorders) | 1 | 0
AUTONOMIC NERVOUS SYSTEM IMBALANCE (Nervous system disorders) | 1 | 0
BALANCE DISORDER (Nervous system disorders) | 1 | 1
BURNING SENSATION (Nervous system disorders) | 1 | 0
CAROTID ARTERY DISEASE (Nervous system disorders) | 2 | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 15 | 9
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 4 | 2
CAUDA EQUINA SYNDROME (Nervous system disorders) | 1 | 0
CENTRAL NERVOUS SYSTEM LESION (Nervous system disorders) | 1 | 0
CEREBELLAR INFARCTION (Nervous system disorders) | 1 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 1 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 20 | 15
CEREBROVASCULAR DISORDER (Nervous system disorders) | 1 | 1
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 1 | 1
COMPLICATED MIGRAINE (Nervous system disorders) | 2 | 0
CONVULSION (Nervous system disorders) | 4 | 2
CUBITAL TUNNEL SYNDROME (Nervous system disorders) | 0 | 1
DEMENTIA (Nervous system disorders) | 0 | 1
DIABETIC NEUROPATHY (Nervous system disorders) | 1 | 1
DIZZINESS (Nervous system disorders) | 58 | 27
DIZZINESS EXERTIONAL (Nervous system disorders) | 2 | 0
DIZZINESS POSTURAL (Nervous system disorders) | 7 | 0
DYSAESTHESIA (Nervous system disorders) | 1 | 0
DYSARTHRIA (Nervous system disorders) | 4 | 0
DYSGEUSIA (Nervous system disorders) | 1 | 0
EMBOLIC STROKE (Nervous system disorders) | 1 | 0
ENCEPHALOPATHY (Nervous system disorders) | 1 | 1
ESSENTIAL TREMOR (Nervous system disorders) | 1 | 0
GUILLAIN-BARRE SYNDROME (Nervous system disorders) | 1 | 0
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 | 1
HAEMORRHAGIC STROKE (Nervous system disorders) | 1 | 0
HEAD DISCOMFORT (Nervous system disorders) | 1 | 0
HEAD TITUBATION (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 28 | 19
HEMIPARESIS (Nervous system disorders) | 1 | 1
HEMIPLEGIC MIGRAINE (Nervous system disorders) | 1 | 0
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
HYPOAESTHESIA (Nervous system disorders) | 13 | 8
HYPOXIC-ISCHAEMIC ENCEPHALOPATHYv (Nervous system disorders) | 2 | 0
IIIRD NERVE PARALYSIS (Nervous system disorders) | 1 | 0
INTENTION TREMOR (Nervous system disorders) | 0 | 1
ISCHAEMIC STROKE (Nervous system disorders) | 6 | 3
LACUNAR INFARCTION (Nervous system disorders) | 1 | 1
LATERAL MEDULLARY SYNDROME (Nervous system disorders) | 1 | 0
LETHARGY (Nervous system disorders) | 2 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 2 | 0
LUMBAR RADICULOPATHY (Nervous system disorders) | 2 | 2
MEMORY IMPAIRMENT (Nervous system disorders) | 6 | 0
MENTAL IMPAIRMENT (Nervous system disorders) | 1 | 0
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 2 | 1
MIGRAINE (Nervous system disorders) | 3 | 1
MYELOMALACIA (Nervous system disorders) | 1 | 0
NERVE COMPRESSION (Nervous system disorders) | 1 | 2
NEURALGIA (Nervous system disorders) | 0 | 1
NEUROLOGICAL SYMPTOM (Nervous system disorders) | 1 | 2
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0
NYSTAGMUS (Nervous system disorders) | 2 | 0
PARAESTHESIA (Nervous system disorders) | 8 | 4
POLYNEUROPATHY ALCOHOLIC (Nervous system disorders) | 1 | 0
POST-TRAUMATIC HEADACHE (Nervous system disorders) | 0 | 2
PRESYNCOPE (Nervous system disorders) | 26 | 8
RADICULITIS (Nervous system disorders) | 1 | 1
RADICULITIS CERVICAL (Nervous system disorders) | 1 | 0
SCIATICA (Nervous system disorders) | 4 | 2
SENSORY DISTURBANCE (Nervous system disorders) | 1 | 0
SOMNOLENCE (Nervous system disorders) | 3 | 0
SPEECH DISORDER (Nervous system disorders) | 0 | 1
SPONDYLITIC MYELOPATHY (Nervous system disorders) | 1 | 0
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 | 1
SUBDURAL HYGROMA (Nervous system disorders) | 2 | 0
SYNCOPE (Nervous system disorders) | 40 | 22
THALAMIC INFARCTION (Nervous system disorders) | 3 | 0
THROMBOTIC STROKE (Nervous system disorders) | 0 | 1
TRANSIENT GLOBAL AMNESIA (Nervous system disorders) | 2 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 17 | 8
TREMOR (Nervous system disorders) | 4 | 2
UNRESPONSIVE TO STIMULI (Nervous system disorders) | 1 | 0
URAEMIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
VERTEBRAL ARTERY OCCLUSION (Nervous system disorders) | 0 | 1
VITH NERVE PARALYSIS (Nervous system disorders) | 2 | 1
ACUTE STRESS DISORDER (Psychiatric disorders) | 0 | 1
ADJUSTMENT DISORDER WITH MIXED DISTURBANCE OF EMOTION AND CONDUCT (Psychiatric disorders) | 0 | 1
AFFECTIVE DISORDER (Psychiatric disorders) | 1 | 0
ALCOHOL ABUSE (Psychiatric disorders) | 1 | 1
ALCOHOL PROBLEM (Psychiatric disorders) | 1 | 0
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 0 | 1
ANXIETY (Psychiatric disorders) | 20 | 7
ANXIETY DISORDER (Psychiatric disorders) | 1 | 0
BIPOLAR DISORDER (Psychiatric disorders) | 0 | 1
BIPOLAR I DISORDER (Psychiatric disorders) | 1 | 0
COMPLETED SUICIDE (Psychiatric disorders) | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 4 | 2
DELIRIUM (Psychiatric disorders) | 1 | 1
DELIRIUM TREMENS (Psychiatric disorders) | 0 | 1
DEPRESSED MOOD (Psychiatric disorders) | 1 | 0
DEPRESSION (Psychiatric disorders) | 17 | 3
DEPRESSION SUICIDAL (Psychiatric disorders) | 1 | 1
HALLUCINATION (Psychiatric disorders) | 0 | 1
HALLUCINATION, VISUAL (Psychiatric disorders) | 0 | 1
INSOMNIA (Psychiatric disorders) | 4 | 3
INTENTIONAL SELF-INJURY (Psychiatric disorders) | 1 | 0
MAJOR DEPRESSION (Psychiatric disorders) | 2 | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 6 | 2
OBSESSIVE-COMPULSIVE DISORDER (Psychiatric disorders) | 0 | 1
PANIC ATTACK (Psychiatric disorders) | 2 | 1
STRESS (Psychiatric disorders) | 1 | 0
SUICIDAL IDEATION (Psychiatric disorders) | 0 | 2
BLADDER DISORDER (Renal and urinary disorders) | 0 | 1
CALCULUS URETERIC (Renal and urinary disorders) | 1 | 3
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 2 | 0
CYSTITIS INTERSTITIAL (Renal and urinary disorders) | 1 | 0
DYSURIA (Renal and urinary disorders) | 4 | 0
HAEMATURIA (Renal and urinary disorders) | 13 | 11
HYDRONEPHROSIS (Renal and urinary disorders) | 2 | 1
HYPERTONIC BLADDER (Renal and urinary disorders) | 1 | 0
MICROALBUMINURIA (Renal and urinary disorders) | 1 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 18 | 10
NOCTURIA (Renal and urinary disorders) | 1 | 0
POLLAKIURIA (Renal and urinary disorders) | 1 | 0
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 1 | 3
RENAL CYST (Renal and urinary disorders) | 4 | 2
RENAL DISORDER (Renal and urinary disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 8 | 5
RENAL FAILURE ACUTE (Renal and urinary disorders) | 17 | 14
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 3 | 5
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 | 2
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 1 | 0
STRESS URINARY INCONTINENCE (Renal and urinary disorders) | 1 | 0
URETHRAL STENOSIS (Renal and urinary disorders) | 1 | 0
URINARY HESITATION (Renal and urinary disorders) | 1 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 2 | 0
URINARY RETENTION (Renal and urinary disorders) | 12 | 3
URINE FLOW DECREASED (Renal and urinary disorders) | 1 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 7 | 5
BREAST CALCIFICATIONS (Reproductive system and breast disorders) | 1 | 0
BREAST MASS (Reproductive system and breast disorders) | 2 | 0
BREAST PAIN (Reproductive system and breast disorders) | 1 | 0
DYSFUNCTIONAL UTERINE BLEEDING (Reproductive system and breast disorders) | 1 | 0
EPIDIDYMAL CYST (Reproductive system and breast disorders) | 0 | 1
FALLOPIAN TUBE CYST (Reproductive system and breast disorders) | 1 | 0
FEMALE GENITAL TRACT FISTULA (Reproductive system and breast disorders) | 1 | 0
HAEMATOSPERMIA (Reproductive system and breast disorders) | 3 | 0
MENORRHAGIA (Reproductive system and breast disorders) | 0 | 2
PELVIC HAEMATOMA (Reproductive system and breast disorders) | 1 | 0
PENILE HAEMORRHAGE (Reproductive system and breast disorders) | 2 | 0
POLYCYSTIC OVARIES (Reproductive system and breast disorders) | 1 | 0
PROSTATITIS (Reproductive system and breast disorders) | 2 | 0
PROSTATOMEGALY (Reproductive system and breast disorders) | 1 | 1
SEXUAL DYSFUNCTION (Reproductive system and breast disorders) | 1 | 0
SPERMATOCELE (Reproductive system and breast disorders) | 1 | 0
TESTICULAR PAIN (Reproductive system and breast disorders) | 1 | 0
UTERINE POLYP (Reproductive system and breast disorders) | 1 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 2 | 1
VULVA CYST (Reproductive system and breast disorders) | 1 | 0
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 4
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 18 | 7
ALLERGIC GRANULOMATOUS ANGIITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 6 | 4
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 2 | 1
BRONCHIAL HYPERREACTIVITY (Respiratory, thoracic and mediastinal disorders) | 0 | 1
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CHOKING (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 35 | 15
COUGH (Respiratory, thoracic and mediastinal disorders) | 21 | 12
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 126 | 55
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 51 | 33
DYSPNOEA PAROXYSMAL NOCTURNAL (Respiratory, thoracic and mediastinal disorders) | 0 | 1
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 26 | 15
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 2 | 5
HYPERVENTILATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 3 | 2
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
MEDIASTINAL MASS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
NASAL POLYPS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
NASAL SEPTUM ULCERATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
NON-CARDIOGENIC PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ORGANISING PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 | 3
ORTHOPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 0
PHARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 9 | 6
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 4 | 2
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 4
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 | 6
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 9 | 7
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 2
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 3 | 2
RESPIRATORY ALKALOSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 2 | 0
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 14 | 8
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 3 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 | 1
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 8 | 6
THROAT TIGHTNESS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
TRACHEAL STENOSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
UPPER RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 2 | 0
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 2 | 1
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 2 | 1
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 3 | 1
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 1
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 1 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 2 | 0
DIABETIC FOOT (Skin and subcutaneous tissue disorders) | 3 | 0
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 | 2
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 3 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 2 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 5 | 1
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 0 | 2
INCREASED TENDENCY TO BRUISE (Skin and subcutaneous tissue disorders) | 9 | 5
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 | 1
LICHENOID KERATOSIS (Skin and subcutaneous tissue disorders) | 1 | 0
LIVEDO RETICULARIS (Skin and subcutaneous tissue disorders) | 1 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 | 1
PRECANCEROUS SKIN LESION (Skin and subcutaneous tissue disorders) | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 4 | 2
PRURITUS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 | 1
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 15 | 8
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 2 | 1
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 2 | 1
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0
SKIN LESION (Skin and subcutaneous tissue disorders) | 2 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 5 | 3
SWELLING FACE (Skin and subcutaneous tissue disorders) | 2 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 4 | 0
AORTIC ANEURYSM REPAIR (Surgical and medical procedures) | 1 | 0
CARDIAC ABLATION (Surgical and medical procedures) | 0 | 1
CARDIAC PACEMAKER BATTERY REPLACEMENT (Surgical and medical procedures) | 0 | 1
CARDIAC PACEMAKER REPLACEMENT (Surgical and medical procedures) | 1 | 0
CHOLECYSTECTOMY (Surgical and medical procedures) | 1 | 1
COLOSTOMY (Surgical and medical procedures) | 0 | 1
CORONARY ARTERY BYPASS (Surgical and medical procedures) | 1 | 0
DENTAL IMPLANTATION (Surgical and medical procedures) | 1 | 0
HERNIA HIATUS REPAIR (Surgical and medical procedures) | 1 | 0
HIP ARTHROPLASTY (Surgical and medical procedures) | 3 | 0
INGUINAL HERNIA REPAIR (Surgical and medical procedures) | 0 | 1
KNEE ARTHROPLASTY (Surgical and medical procedures) | 1 | 0
LEG AMPUTATION (Surgical and medical procedures) | 0 | 1
MEDICAL DEVICE REMOVAL (Surgical and medical procedures) | 0 | 1
NEPHRECTOMY (Surgical and medical procedures) | 1 | 0
SINUS OPERATION (Surgical and medical procedures) | 1 | 0
SPINAL FUSION SURGERY (Surgical and medical procedures) | 1 | 0
TENDON OPERATION (Surgical and medical procedures) | 0 | 1
THERAPY CESSATION (Surgical and medical procedures) | 1 | 0
TONSILLECTOMY (Surgical and medical procedures) | 0 | 1
TOOTH EXTRACTION (Surgical and medical procedures) | 0 | 1
TRANSURETHRAL PROSTATECTOMY (Surgical and medical procedures) | 0 | 1
ACCELERATED HYPERTENSION (Vascular disorders) | 4 | 1
AORTIC ANEURYSM (Vascular disorders) | 8 | 3
AORTIC DISSECTION (Vascular disorders) | 0 | 1
AORTIC INTRAMURAL HAEMATOMA (Vascular disorders) | 1 | 1
AORTIC STENOSIS (Vascular disorders) | 4 | 5
ARTERIAL SPASM (Vascular disorders) | 1 | 0
ARTERIOSCLEROSIS (Vascular disorders) | 0 | 1
ARTERIOVENOUS FISTULA (Vascular disorders) | 1 | 0
BLEEDING VARICOSE VEIN (Vascular disorders) | 1 | 0
BLOOD PRESSURE FLUCTUATION (Vascular disorders) | 0 | 1
BLOOD PRESSURE INADEQUATELY CONTROLLED (Vascular disorders) | 1 | 0
CIRCULATORY COLLAPSE (Vascular disorders) | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 12 | 8
ESSENTIAL HYPERTENSION (Vascular disorders) | 1 | 1
FEMORAL ARTERIAL STENOSIS (Vascular disorders) | 2 | 1
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 0 | 1
FLUSHING (Vascular disorders) | 0 | 1
HAEMATOMA (Vascular disorders) | 8 | 1
HAEMORRHAGE (Vascular disorders) | 2 | 1
HOT FLUSH (Vascular disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 60 | 24
HYPERTENSIVE CRISIS (Vascular disorders) | 7 | 7
HYPOTENSION (Vascular disorders) | 38 | 13
ILIAC ARTERY OCCLUSION (Vascular disorders) | 1 | 0
ILIAC ARTERY STENOSIS (Vascular disorders) | 1 | 1
INTERMITTENT CLAUDICATION (Vascular disorders) | 14 | 10
LABILE HYPERTENSION (Vascular disorders) | 1 | 0
MALIGNANT HYPERTENSION (Vascular disorders) | 1 | 0
ORTHOSTATIC HYPERTENSION (Vascular disorders) | 1 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 8 | 3
PALLOR (Vascular disorders) | 1 | 0
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 5 | 10
PERIPHERAL COLDNESS (Vascular disorders) | 2 | 0
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 | 1
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 8 | 6
POOR PERIPHERAL CIRCULATION (Vascular disorders) | 1 | 0
RAYNAUD'S PHENOMENON (Vascular disorders) | 1 | 0
REPERFUSION INJURY (Vascular disorders) | 5 | 2
SUBCLAVIAN ARTERY OCCLUSION (Vascular disorders) | 1 | 0
SUBCLAVIAN ARTERY STENOSIS (Vascular disorders) | 1 | 0
SUBCLAVIAN STEAL SYNDROME (Vascular disorders) | 1 | 0
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 1 | 1
THROMBOSIS (Vascular disorders) | 3 | 0
VARICOSE VEIN (Vascular disorders) | 1 | 0
VASOSPASM (Vascular disorders) | 1 | 0
VENOUS INSUFFICIENCY (Vascular disorders) | 1 | 0
WEGENER'S GRANULOMATOSIS (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less